# 1.0 Title Page

# **Statistical Analysis Plan**

# **Study M15-555**

A Phase 3, Randomized, Double-Blind Study
Comparing Upadacitinib Monotherapy to
Methotrexate (MTX) in Subjects with Moderately to
Severely Active Rheumatoid Arthritis with
Inadequate Response to MTX

Date: 17 Dec 2020

**Version 3.0** 

# **Table of Contents**

| 1.0 | Title Page | 1 |
|---|---|---|
| 2.0 | Introduction | <mark>7</mark> |
| 3.0 | Study Objectives, Design and Procedures | <mark>7</mark> |
| 3.1 | Study Objectives | 7 |
| 3.2 | Overall Study Design and Plan | 7 |
| 3.3 | Sample Size | 14 |
| 3.4 | Interim Analysis and Data Base Lock | 15 |
| 3.5 | Data Monitoring Committee (DMC) Activities | 15 |
| 4.0 | Analysis Populations and Analysis Windows | 15 |
| 4.1 | Analysis Populations | 15 |
| 4.2 | Analysis Windows | 16 |
| 5.0 | Demographics, Baseline Characteristics, Medical History, and Previous/Concomitant Medications | 18 |
| 5.1 | Demographic and Baseline Characteristics | |
| 5.2 | Medical History | |
| 5.3 | Previous Treatment and Concomitant Medications | |
| 5.4 | Protocol Deviations | 22 |
| 6.0 | Patient Disposition | 22 |
| 7.0 | Study Drug Exposure and Compliance | 24 |
| 7.1 | Study Drug Exposure | |
| 7.2 | Compliance | 26 |
| 8.0 | Efficacy Analysis | 26 |
| 8.1 | General Considerations | 26 |
| 8.1.1 | Efficacy Analysis at Different Phases of the Study | 26 |
| 8.1.2 | Definition of Missing Data Imputation | 27 |
| 8.2 | Efficacy Analysis for Period 1 | 30 |
| 8.2.1 | Primary Efficacy Analysis | 30 |
| 8.2.2 | Sensitivity Analysis of Primary Efficacy Variables | 30 |
| 8.2.3 | Key Secondary Efficacy Analyses | 30 |
| 8.2.4 | Exploratory Efficacy Analyses | 32 |
| 8.2.5 | Handling of Multiplicity | 33 |

# Upadacitinib M15-555 – Statistical Analysis Plan Version 3.0 – 17 Dec 2020

| 8.2.6 | Efficacy Subgroup Analysis | 36 |
|---|---|---|
| 8.2.7 | Summary of Efficacy Analysis for Period 1 | 37 |
| 8.3 | Long-Term Efficacy Analyses | |
| 8.4 | Efficacy Variables Definitions and Conventions | 42 |
| 8.4.1 | ACR Criteria | 42 |
| 8.4.2 | Joint Evaluation | 45 |
| 8.4.3 | Patient's Global Assessment of Disease Activity Visual Analog Scale (VAS) | 46 |
| 8.4.4 | Physician's Global Assessment of Disease Activity Visual Analog Scale (VAS) | 47 |
| 8.4.5 | Patient's Global Assessment of Pain | 47 |
| 8.4.6 | Disease Activity Score (DAS28) | 47 |
| 8.4.7 | Simplified Disease Activity Index (SDAI) | 48 |
| 8.4.8 | Clinical Disease Activity Index (CDAI) | 48 |
| 8.4.9 | Clinical Remission (CR) and Low Disease Activity (LDA) | 49 |
| 8.4.10 | ACR/EULAR Boolean Remission | 49 |
| 8.4.11 | Disability Index of Health Assessment Questionnaire (HAQ-DI) | 49 |
| 8.4.12 | EuroQoL-5D (EQ-5D-5L) | 50 |
| 8.4.13 | Form SF-36v2 | 50 |
| 9.0 | Safety Analysis | <b>51</b> |
| 9.1 | General Considerations | 51 |
| 9.2 | Analysis of Adverse Events | 53 |
| 9.2.1 | Analysis of Adverse Events for Period 1 | |
| 9.2.1.1 | Adverse Events Overview | 53 |
| 9.2.1.2 | Adverse Events by System Organ Class and Preferred Term | 54 |
| 9.2.1.3 | TEAEs by Maximum Severity | 55 |
| 9.2.1.4 | TEAEs by Relationship | 55 |
| 9.2.1.5 | Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term | 56 |
| 9.2.1.6 | Adverse Events of Special Interest | |
| 9.2.2 | Analysis of Long-Term Adverse Event Rates | |

# Upadacitinib M15-555 – Statistical Analysis Plan Version 3.0 – 17 Dec 2020

| Assessment of Potentially Clinical Significant Laboratory Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations Analysis of Vital Signs Variables and Criteria Defining Abnormality Analysis of Vital Signs for Period 1 Analysis of Long-Term Vital Signs Summary of Changes Summary of Changes between the Previous Version and the Current Version Version History Appendix | 6566666868697070 |
|---|---|
| Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations Analysis of Vital Signs Variables and Criteria Defining Abnormality Analysis of Vital Signs for Period 1 Analysis of Long-Term Vital Signs Summary of Changes Summary of Changes between the Previous Version and the Current Version | 65666668686970 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations Analysis of Vital Signs Variables and Criteria Defining Abnormality Analysis of Vital Signs for Period 1 Analysis of Long-Term Vital Signs Summary of Changes Summary of Changes between the Previous Version and the | 65<br>66<br>66<br>68<br>68<br>68 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations Analysis of Vital Signs Variables and Criteria Defining Abnormality Analysis of Vital Signs for Period 1 Analysis of Long-Term Vital Signs Summary of Changes | 65<br>66<br>66<br>67<br>68<br>68 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations Analysis of Vital Signs Variables and Criteria Defining Abnormality Analysis of Vital Signs for Period 1 Analysis of Long-Term Vital Signs | 65<br>66<br>66<br>67<br>68<br>68 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations Analysis of Vital Signs Variables and Criteria Defining Abnormality Analysis of Vital Signs for Period 1 | 65<br>66<br>66<br>67<br>68<br>68 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations Analysis of Vital Signs Variables and Criteria Defining Abnormality | 65<br>66<br>66<br>67<br>68 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations Analysis of Vital Signs | 65<br>66<br>66<br>67 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values Assessment of Liver Elevations | 65<br>66<br>66<br>66 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables Assessment of Potentially Clinical Significant Laboratory Values | 65<br>66<br>66 |
| Variables Assessment of Liver Elevations Analysis of Long-Term Laboratory Data Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables | 65<br>66 |
| Variables | 65 |
| Variables | 65 |
| Variables | |
| | 64 |
| Assessment of Shift from Baseline in Clinical Laboratory Variables | 64 |
| Assessment of Mean Change from Baseline and Percentage Change from Baseline in Clinical Laboratory Variables | 63 |
| Analysis of Laboratory Data for Period 1 | 63 |
| Analysis of Laboratory Data | 61 |
| Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation | 61 |
| Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure | 60 |
| Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT | |
| Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure | 58 |
| | Study Drug Exposure Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation Analysis of Laboratory Data Variables and Units Analysis of Laboratory Data for Period 1 Assessment of Mean Change from Baseline and Percentage Change from Baseline in Clinical Laboratory Assessment of Shift from Baseline in Clinical Laboratory |



# **List of Tables**

| Table 1. | Analysis Windows for Efficacy Analysis by Week 14 (for ACR Components and Morning Stiffness) and Safety Analysis by Week 14 (for Labs and Vital Signs) |
|---|---|
| Table 2. | Analysis Windows for Efficacy Analysis by Week 14 (for EQ-5D-5L and SF-36) |
| Table 3. | Analysis Windows for Safety Analysis by Week 14 (for IgG and IgM) |
| Table 4. | Subgroups for Efficacy Analysis |
| Table 5. | Summary of Efficacy Variables and Corresponding Analyses for Efficacy Analysis in Period 1 |
| Table 6. | Summary of Efficacy Variables and Corresponding Analyses for Long-Term Efficacy Analysis |
| Table 7. | Anatomical Joints Assessed for Calculation of Tender and Swollen Joint Counts (TJC68 and SJC66) |
| Table 8. | Anatomical Joints for DAS28 (CRP) Calculation48 |
| Table 9. | AESI for Upadacitinib with SMQs/CMQs/PTs Searches56 |
| Table 10. | List of Laboratory Variables |
| Table 11. | Criteria for Potentially Clinically Significant Vital Sign Findings68 |
| Table 12. | SAP Version History Summary |
| List of Figu | res |
| Figure 1. | Period 1 Study Design |
| Figure 2. | Period 2 Study Design |
| Figure 3. | Graphical Multiple Testing Procedure for US/FDA Regulatory Purposes |
| Figure 4. | Graphical Multiple Testing Procedure for EU/EMA Regulatory Purposes |
| List of Appe | endices |
| Appendix A. Appendix B. | OMERACT Criteria |



| M15-555 – Statistical Analysis l | Plan |
|----------------------------------|------|
| Version 3.0 – 17 Dec 2020 | |

| Appendix C. | Statistical Analysis to Account for Impact of COVID-19 |
|-------------|--------------------------------------------------------|
| | Pandemic 86 |



#### 2.0 Introduction

This statistical analysis plan (SAP) describes the statistical analyses to be completed by the Data and Statistical Science Department for Upadacitinib Study M15-555. It provides details to further elaborate statistical methods as outlined in the protocol.

Pharmacokinetic and exploratory biomarker analyses will be performed separately and the corresponding analysis plan is documented separately. Unless noted otherwise, all analyses will be performed using SAS version 9.2 or later (SAS Institute Inc., Cary, NC 27513) under the UNIX operating system.

### 3.0 Study Objectives, Design and Procedures

#### 3.1 Study Objectives

#### Period 1

To compare the safety and efficacy (signs and symptoms) of Upadacitinib 30 mg once daily (QD) alone and 15 mg QD alone versus continuing methotrexate (MTX) alone in MTX-inadequate response (MTX-IR) subjects with moderately to severely active rheumatoid arthritis (RA).

#### Period 2

To evaluate the long-term safety, tolerability, and efficacy of Upadacitinib 30 mg QD and 15 mg QD in subjects with RA who have completed Period 1.

#### 3.2 Overall Study Design and Plan

This is a Phase 3 multicenter study that includes two periods. Period 1 is a 14-week, randomized, double-blind, parallel-group, controlled period designed to compare the safety and efficacy of Upadacitinib 30 mg QD alone and 15 mg QD alone versus continuing MTX alone for the treatment of signs and symptoms of RA in subjects with moderately to severely active RA despite stable doses of MTX (inadequate response to MTX). Period 2 is a blinded long-term extension period to evaluate the long-term safety,



tolerability, and efficacy of Upadacitinib 30 mg QD and 15 mg QD in subjects with RA who have completed Period 1. Starting with Amendment 5, all subjects will receive openlabel upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD.

The study is designed to enroll 600 subjects at approximately 175 study centers worldwide to meet scientific and regulatory objectives without enrolling an undue number of subjects in alignment with ethical considerations. Therefore, if the target number of subjects has been enrolled, there is a possibility that additional subjects in screening may not be enrolled.

The study duration includes a 35-day screening period; a 14-week randomized, double-blind, parallel-group, controlled treatment period (Period 1); a 246-week blinded extension period (Period 2); and a 30-day follow-up visit.

Subjects who meet eligibility criteria will be randomized in a 2:2:1:1 ratio to one of four treatment groups:

- Group 1: Upadacitinib 30 mg QD (N = 200) (Period 1) → Upadacitinib 30 mg QD (Period 2)
- Group 2: Upadacitinib 15 mg QD (N = 200) (Period 1) → Upadacitinib 15 mg QD (Period 2)
- Group 3: MTX (N = 100) (Period 1) → Upadacitinib 30 mg QD (Period 2)
- Group 4: MTX (N = 100) (Period 1) → Upadacitinib 15 mg QD (Period 2)

Randomization is stratified by geographic region.

Prior to enrollment subjects must have been receiving oral or parenteral MTX therapy  $\geq 3$  months and on a stable dose [15 to 25 mg/week; or  $\geq 10$  mg/week in subjects who are intolerant of MTX at doses  $\geq 12.5$  mg/week (For subjects in Japan: the minimum dose is 10 mg/week; or 7.5 mg/week in subjects who are intolerant of MTX at doses  $\geq 10$  mg/week)] for at least 4 weeks. No MTX washout is needed prior to randomization. Each subject will be instructed to take a required number of capsules once weekly (MTX)



and/or matching placebo) based on prior dose of MTX and 1 tablet once daily (Upadacitinib or matching placebo) to maintain blinding. MTX and matching placebo will be distributed as active MTX or placebo tablets over-encapsulated into identical capsules to in blister packs, to provide the correct total dose for each individual subject and to maintain blinding during Period 1.

All subjects will start on their blinded Upadacitinib (30 mg QD, 15 mg QD or Placebo QD) dose at Baseline. Also, starting at Baseline, all subjects will discontinue their current MTX treatment and start their blinded MTX treatment. Subjects will be given oral MTX in a blinded manner (7.5 to 25 mg/week or placebo) based on the subject's prior stable dose of MTX and per protocol instructions. For all other doses of MTX, subjects will be assigned to blinded MTX based on their current stable MTX dose at study entry. In addition, all subjects should take a dietary supplement of folic acid (or equivalent) throughout Period 1 participation; while in Period 2 (starting at Week 26) it should only be taken if MTX is given as background medication. Folic acid dosing and timing of regimen should be followed according to Investigator's instructions.

Subjects who complete the Week 14 visit (end of Period 1) will enter the blinded long-term extension portion of the study, Period 2 (246 weeks). Subjects who are assigned to Upadacitinib treatment groups in Period 1 will continue to receive Upadacitinib 30 mg QD or 15 mg QD per original randomization assignment in a blinded manner. Subjects who are assigned to MTX treatment group in Period 1 will discontinue MTX and receive Upadacitinib 30 mg QD or 15 mg QD in a blinded fashion per their prespecified randomization assignments. Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD.

In Period 2, subjects who do not achieve LDA as defined by CDAI  $\leq$  10 at Week 26 should have background medication(s) adjusted or initiated as rescue after assessments for Week 26 have been completed.

An unblinded analysis will be conducted after all subjects have completed Period 1 (Week 14). Study sites and subjects will remain blinded for the duration of the study (Period 1 and Period 2).

Study design schematics of Period 1 and Period 2 are shown in Figure 1 and Figure 2, respectively.

**Screening Period** PERIOD 1: Follow-Up Period (Up to 35 days) (≈ 30 days)\* 14-Week, Randomized, Double-Blind, Treatment Period ABT-494 15 MG QD Adults with n=200 Randomization 2:2:1:1 moderately to severely active ABT-494 30 MG QD RA who have n=200 had an inadequate MTX response to n=100 MTX (no washout MTX required) n=100 Baseline W2 W4 W8 W14

Figure 1. Period 1 Study Design

MTX = methotrexate; n = number; QD = once daily; RA = rheumatoid arthritis; W = week

<sup>\*</sup> The follow-up period is only for subjects who do not enter Period 2.

PERIOD 2: End of Period 1 246-Week Blinded Extension Period (≈ 30 days) ABT-494 15 MG QD **ABT-494 15 MG QD** ABT-494 30 MG QD Amendment 5 ABT-494 15 MG QD MTX **ABT-494 15 MG QD** MTX Amendment 5 ABT-494 30 MG QD ABT-494 15 MG QD W14 W20 W26 W36 W48 W240 (and every 12 W260 weeks) Starting at Week 26, initiation of or change in csDMARDs is allowed

Figure 2. Period 2 Study Design

 $csDMARD = conventional \ synthetic \ disease \ modifying \ anti-rheumatic \ drug; \ MTX = methotrexate; \ QD = once \ daily; \ RA = rheumatoid \ arthritis; \ W = week$ 

Note: Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD.

#### **Screening Period**

Within 35 days prior to the Baseline Visit, subjects will receive a full explanation of the study design and study procedures, provide a written informed consent, and undergo the screening procedures outlined in the protocol. Lab values can be re-tested once during the screening period. If the re-tested lab value(s) remain(s) exclusionary, the subject will be considered a screen failure with no additional re-screening possible. Redrawing samples if initial samples were unable to be analyzed would not count as a retest since initial result was never obtained.

Subjects that initially screen fail for the study are permitted to re-screen once following re-consent. Lab values can be re-tested once during the re-screening period. For



additional re-screenings, AbbVie Therapeutic Area Medical Director approval is required. All screening procedures with the possible exceptions noted below will be repeated during re-screening. The subject must meet all the inclusion and none of the exclusion criteria at the time of re-screening in order to qualify for the study. There is no minimum period of time a subject must wait to re-screen for the study. If the subject had a complete initial screening evaluation including the assessment of an Interferon-Gamma Release Assay (IGRA; QuantiFERON Tuberculosis [TB] Gold In Tube test) or a purified protein derivative (PPD) test (or equivalent), or chest x-ray and electrocardiogram (ECG), these tests will not be required to be repeated for re-screening provided the conditions noted in protocol are met and no more than 90 days have passed.

#### Period 1 (14-Week Randomized, Double-Blind Treatment Period)

Period 1 will begin at the Baseline Visit (Day 1) and will end at the Week 14 Visit. At the Baseline Visit, subjects who meet all the inclusion criteria and none of the exclusion criteria described in the protocol will be enrolled into the study and randomized to double-blind treatment. During this period of the study, subjects will visit the study site at Weeks 2, 4, 8, and 14.  $A \pm 3$  day window is permitted around scheduled study visits. The last dose of the daily study drug tablets in Period 1 is taken the day prior to the Week 14 visit.

#### Period 2 (Blinded Long-Term Extension Period [246 Weeks])

Period 2 will begin at the Week 14 Visit after all assessments have been completed. During Period 2, subjects will have a study visit at Weeks 20, 26, 36, 48, and every 12 weeks through Week 240 and Week 260. A  $\pm$  7 day window is permitted around scheduled study visits. Starting at Week 26 and thereafter, at least 20% improvement in BOTH TJC AND SJC is required to remain on study drug. Anyone who does not fulfill this criterion at 2 consecutive visits (starting at Week 26) must be discontinued from study drug.

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD.



# <u>Discontinuation of Study Drug and Continuation of Study Participation (Period 1 and Period 2)</u>

Subjects may discontinue study drug treatment, but may choose to continue to participate in the study. Subjects who prematurely discontinue study drug should complete a Premature Discontinuation visit (PD visit) as soon as possible, preferably within 2 weeks. To minimize missing data for efficacy and safety assessments, subjects who prematurely discontinue study drug treatment should continue to be followed for all regularly scheduled visits as outlined in the protocol, unless subjects have decided to discontinue study participation entirely (withdrawal of informed consent). Subjects should be advised on the continued scientific importance of their data even if they discontinue treatment with study drug early. Following discontinuation of study drug, the subject should be treated in accordance with the investigator's best clinical judgment irrespective of whether the subject decides to continue participation in the study. As the subject has discontinued study drug, all rescue- and efficacy-driven discontinuation criteria no longer apply. This includes the 20% TJC/SJC calculations at Week 26 and visits thereafter, as well as the CDAI calculation at Week 26, if applicable. If at any point a subject withdraw consent following discontinuation of study drug and no longer wants to provide assessments, a second PD visit is not required.

# <u>Premature Discontinuation of Study (Withdrawal of Informed Consent) (Period 1 and Period 2)</u>

Subjects may withdraw from the study completely (withdrawal of informed consent) for any reason at any time. If a subject prematurely discontinues study drug treatment AND study participation (withdrawal of informed consent), the procedures outlined for the Premature Discontinuation visit (PD visit) should be completed as soon as possible, preferably within 2 weeks of study drug discontinuation. In addition, if the subject is willing, a 30-day follow-up visit (or phone call, if a visit is not possible) may occur to determine the status of any ongoing AEs/SAEs or the occurrence of any new AEs/SAEs.



#### Follow-Up Visit

A Follow-Up Visit will occur approximately 30 days after the last dose of study drug to obtain information on any new or ongoing AE/SAEs, and to collect vital signs and clinical laboratory tests.

Subjects will complete the Follow-Up Visit when they have either:

- Completed the last visit of Period 1 (Week 14), but decided not to participate in the extension Period 2; OR
- Completed the last visit of Period 2; OR
- Prematurely discontinued study drug and study participation (withdrawal of consent). If a PD visit has already occurred then the 30 day follow-up visit may be a telephone call if a site visit is not possible. Vital signs and laboratory test may not be required. The Follow-Up Visit is not applicable for subjects who discontinued study drug and continued study participation and completed at least one study visit at least approximately 30 days after last dose.

#### 3.3 Sample Size

The planned total sample size of 600 for this study provides at least 90% power to detect a 21% difference in ACR20 response rate (assuming an ACR20 response rate of 37% in the MTX group), as well as at least 90% power to detect a 22% difference in LDA response rate based on DAS28 (CRP) criteria (assuming an LDA response rate of 15% in the MTX group), at two-sided  $\alpha = 0.025$  and accounting for 10% dropout rate. This sample size will also provide at least 90% power for most of the key secondary endpoints, including change from baseline in DAS28 (CRP), ACR50, change from baseline in HAQ-DI, CR based on DAS28 (CRP), and change from baseline in SF-36 PCS at two-sided significance level of 0.025 and accounting for a 10% dropout rate.



#### 3.4 Interim Analysis and Data Base Lock

An unblinded analysis will be conducted after all subjects have completed Period 1 (Week 14). Study sites and subjects will remain blinded for the duration of the study (Periods 1 and 2).

#### 3.5 Data Monitoring Committee (DMC) Activities

An independent external Data Monitoring Committee (DMC) is used to review unblinded safety data at regular intervals during the conduct of the study. The DMC will provide recommendation to an AbbVie Point of Contact on whether to continue, modify, or terminate studies after each review. When needed, high level unblinded efficacy data may also be requested by the DMC and be reviewed so that the DMC can assess benefit: risk of any emerging safety differences.

#### 4.0 Analysis Populations and Analysis Windows

### 4.1 Analysis Populations

#### Full Analysis Set (FAS)

The Full Analysis Set (FAS) includes all randomized subjects who received at least one dose of study drug. The FAS will be used for all efficacy and baseline analyses.

#### Per Protocol Analysis Set

The Per Protocol Analysis Set represents a subset of the FAS and consists of all FAS subjects who did not meet any major protocol deviations during Period 1 of the study. Additional analysis of the primary efficacy endpoint will be conducted on the Per Protocol analysis set, in order to evaluate the impact of major protocol deviations.

Major protocol deviations (ICH deviation and other clinically significant non-ICH deviation) will be identified prior to database lock.



#### Safety Analysis Set

The Safety Analysis Set consists of all subjects who received at least one dose of study drug. For the Safety Analysis Set, subjects are assigned to a treatment group based on the "as treated" treatment group, regardless of the treatment randomized. The "as treated" is determined by the treatment the subject received during the majority of the subject's drug exposure time in the analysis period.

#### 4.2 Analysis Windows

#### **Definition of Study Days (Days Relative to the First Dose of Study Drug)**

Study Days are calculated for each collection date relative to the date of the first dose of study drug. It is defined as the number of days between the date of the first dose of study drug and the collection date. Study days are negative values when the collection date of interest is prior to the first study drug dose date. Study days are positive values when the collection date of interest is on or after the first study drug dose date. The day of the first dose of study drug is defined as Study Day 1, while the day prior to the first study drug dose is defined as Study Day –1 (there is no Study Day 0). Study days are used to map actual study visits to the protocol-specified study visits.

#### **Definition of Analysis Windows**

The following rules will be applied to assign actual subject visits to protocol-specified visits. For each protocol-specified study visit, a target study day will be identified to represent the corresponding visit along with a window around the target day. Windows will be selected in a non-overlapping fashion so that a collection date does not fall into multiple visit windows. If a subject has two or more actual visits in one visit window, the visit closest to the target day will be used for analysis. If two visits are equidistant from the target day, then the later visit will be used for analysis.

The visit window and the target study day for each protocol-specified visit in Period are displayed in Table 1, Table 2, and Table 3 (depending on the different visit schedules of

different endpoints). Visit windows for protocol-specified visits in Period 2 are defined similarly.

Table 1. Analysis Windows for Efficacy Analysis by Week 14 (for ACR Components and Morning Stiffness) and Safety Analysis by Week 14 (for Labs and Vital Signs)

| Protocol Specifie<br>Visit Week | d<br>Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | -99 | 1 a | 1 |
| 2 | 2 | 15 | 22 |
| 4 | 23 | 29 | 43 |
| 8 | 44 | 57 | 78 |
| 14 | 79 | 99 | min (119, first dose date from<br>Week 14 dispensed kit) |

a. Day of first dose of study drug.

Table 2. Analysis Windows for Efficacy Analysis by Week 14 (for EQ-5D-5L and SF-36)

| Protocol Specified<br>Visit Week | d<br>Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | -99 | 1 <sup>a</sup> | 1 |
| 4 | 2 | 29 | 64 |
| 14 | 65 | 99 | min (133, first dose date from<br>Week 14 dispensed kit) |

a. Day of first dose of study drug.

Table 3. Analysis Windows for Safety Analysis by Week 14 (for IgG and IgM)

| Protocol Specified<br>Visit Week | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | -99 | 1ª | 1 |
| 14 | 2 | 99 | min (196, first dose date from Week 14 dispensed kit) |

a. Day of first dose of study drug.

# 5.0 Demographics, Baseline Characteristics, Medical History, and Previous/Concomitant Medications

#### 5.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics information will be collected at the Baseline visit of the study and will be summarized for the FAS. The number of observations, mean, standard deviation, median, minimum and maximum will be summarized for continuous variables. Categorical or discrete variables will be summarized via frequencies and percentages. Summary statistics will be computed for each treatment group and overall.

#### **Main Demographic and Baseline Characteristics**

- Sex (male, female)
- Age (years)
- Age Categories ( $< 40, [40, 65], \ge 65 \text{ years}$ )
- Race (White, Black or African American, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Asian, Other)
- Geographic Region (North America, South/Central America, Western Europe, Eastern Europe, Asia, Other)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Weight (kg)
- Weight Categories ( $< 60 \text{ kg}, \ge 60 \text{ kg}$ )
- Height (cm)
- Body Mass Index (BMI) (kg/m<sup>2</sup>)
- Body Mass Index (BMI) Category (kg/m<sup>2</sup>) (BMI  $\leq$  25, BMI  $\geq$  25)

#### **RA Medical History and Characteristics**

- Duration of RA Symptoms in years
- Duration of RA Diagnosis in years
- Duration of RA Categories ( $< 5 \text{ year}, \ge 5 \text{ year}$ )



- Duration of prior methotrexate therapy
- Prior Methotrexate dose
- Corticosteroids use at baseline (yes, no)
- Oral steroid dosing (prednisone equivalent) at baseline

#### ACR and/or DAS Components at Baseline

- Tender joint count (TJC68) defined as the number of tender joints out of 68 assessed joints
- Swollen joint count (SJC66) defined as the number of swollen joints out of 66 assessed joints
- Tender joint count (TJC28) defined as the number of tender joints out of 28 assessed joints used for DAS28 calculation
- Swollen joint count (SJC28) defined as the number of swollen joints out of 28 assessed joints used for DAS28 calculation
- Physician's global assessment of disease activity (mm on a 100-mm horizontal visual analogue scale [VAS])
- Patient's assessment of pain within last week (mm on a 100-mm horizontal (VAS)
- Patient's global assessment of disease activity within last 24 hours (mm on a 100-mm horizontal VAS)
- Health Assessment Questionnaire Disability Index of the (HAQ DI) (range: 0 to 3)
- High sensitivity C-reactive protein (hsCRP) (mg/L)

#### Other Baseline RA Disease Characteristics

- Anti-cyclic citrulliated peptide (Anti-CCP) (units)
- Anti-CCP status: Positive or Negative
- Rheumatoid Factor (RF) (units)
- Rheumatoid Factor (RF) status: Positive or Negative
- RF and Anti-CCP status: at least one positive or double negative

# Upadacitinib M15-555 – Statistical Analysis Plan Version 3.0 – 17 Dec 2020

- RF and Anti-CCP status: at least one negative or double positive
- DAS28 [hsCRP]
- DAS28 [ESR]
- DAS28 Categories:
  - DAS28 > 5.1 (Severe Disease Activity)
  - o DAS28 ≤ 5.1
- Clinical Disease Activity Index (CDAI)
- CDAI categories:
  - CDAI > 22 (Severe Disease Activity)
  - $\circ$  CDAI  $\leq$  22
- Simplified Disease Activity Index (SDAI)
- SDAI categories:
  - o SDAI > 26 (Severe Disease Activity)
  - $\circ$  SDAI  $\leq 26$

#### **Patient Report Outcomes at Baseline**

- Morning stiffness (severity and duration)
- EQ-5D-5L
- 36-Item Short Form Health Survey (SF-36) Version 2: physical component summary, mental component summary and the 8 sub-domain scores

#### **Clinical Tests at Screening**

- Chest x-ray
- Tuberculin PPD skin test, QuantiFERON TB Gold test
- Serum pregnancy test
- ECG

#### **Immunization History**

• BCG immunization



- Herpes Zoster immunization
- Hepatitis B immunization

#### **Tobacco/Nicotine and Alcohol Use**

- Tobacco/Nicotine Use [user, ex-user, non-user, unknown]
- Alcohol Use [drinker, ex-drinker, non-drinker, unknown]

#### 5.2 Medical History

Medical history data will be summarized and presented for FAS population using body systems and conditions/diagnoses as captured on the CRF. The body systems will be presented in alphabetical order and the conditions/diagnoses will be presented in alphabetical order within each body system. The number and percentage of subjects with a particular condition/diagnosis will be summarized for each randomized treatment group as well as overall. Subjects reporting more than one condition/diagnosis within a body system will be counted only once for that body system. No statistical comparison will be performed for medical history reporting.

#### 5.3 Previous Treatment and Concomitant Medications

Prior and concomitant medications will be summarized by each randomized treatment group as well as overall for FAS. Prior medications are those medications taken prior to the first dose of study drug. This includes medications with a start date before the first study drug administration date, regardless of the end date of these medications. Medications taken on the day of the first dose of study drug are not counted as prior medications. Concomitant medications are those medications, other than study drug, taken after the first dose of study drug and within 7 day of the last dose of study drug. This includes medications with a start date between first study drug administration and last study drug administration + 7 day, as well as, medications with a start date prior to first dose of study drug and which are ongoing after first dose of study drug. Medications taken on the day of the first dose of study drug are counted as concomitant medications.



The number and percentage of subjects who received a prior medication and the number and percentage of subjects who received a concomitant medication will be tabulated separately by the generic name assigned by the most current version of the World Health Organization (WHO) Drug Dictionary.

#### 5.4 Protocol Deviations

Protocol deviations based on ICH deviation criteria are categorized as follows:

- Those who entered the study even though they did not satisfy the entry criteria
- Those who developed withdrawal criteria during the study and were not withdrawn
- Those who received the wrong treatment or incorrect dose, and
- Those who received an excluded or prohibited concomitant medication.

The protocol deviations listed above and other significant protocol deviations will be summarized and listed by treatment group.

# 6.0 Patient Disposition

The following will be summarized by randomized treatment group as well as overall:

- number of subjects randomized,
- number of subjects included in key analysis populations (Full Analysis Set and Per Protocol Analysis Set for primary efficacy analysis, Safety Analysis Set for Period 1),
- number of subjects who completed Period 1 study participation,
- number of subjects who entered Period 2,
- number of subjects on-going in Period 2 (if applicable),
- number of subjects who completed overall study (Period 1 and Period 2) participation.

This summary will be repeated by site.



Premature discontinuation details will be further summarized separately for Period 1 and Period 2 as follows.

#### Period 1

The number and percentage of subjects completed Period 1 and prematurely discontinued in Period 1 will be summarized by randomized treatment group, separately by study drug and study participation completion/discontinuation, with the primary reason for discontinuation collected from CRF by the following categories:

- Adverse event (AE)
- Withdrew consent
- Lost to follow-up
- Lack of efficacy
- Other.

Subjects may have more than one reason for discontinuing, but only the primary reason will be summarized.

In addition, the number and percentage of subjects enrolled in Period 2 will also be summarized by randomized treatment group.

#### Period 2

Period 2 patient dispositions and reason for discontinuation will be summarized for overall and by treatment regimen when entering Period 2 defined as follows:

- 1. Upadacitinib 15 mg QD
- 2. Upadacitinib 30 mg QD

Among the subjects who entered Period 2 participation (regardless of whether subject prematurely discontinued study drug in Period 1), the number and percentage of subjects completed, on-going (if applicable), and prematurely discontinued study participation in



Period 2 will be summarized. Among the subjects who entered Period 2 upon completion of study drug in Period 1, the number and percentage of subjects completed, on-going (if applicable), and prematurely discontinued study drug in Period 2 will be summarized.

For subjects who prematurely discontinued study drug or study participation, the primary reason as well as all reasons for discontinuation will be summarized by the following categories (as collected in CRF):

- Adverse event (AE)
- Withdrew consent
- Lost to follow-up
- Lack of efficacy
- Other.

#### Summary of Dose Switch from Upadacitinib 30 mg QD to 15 mg QD

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD. The visit at which dose switch occurs could be different for each subject. For subjects on upadacitinib 30 mg QD in Period 2, the number and percentage of subjects switching to upadacitinib 15 mg QD at each visit will be summarized.

# 7.0 Study Drug Exposure and Compliance

# 7.1 Study Drug Exposure

The duration of exposure to study drug will be summarized for the safety analysis set by the following groups.

#### 1. MTX



#### 2. Upadacitinib 15 mg QD

This includes Upadacitinib 15 mg QD exposure from subjects starting on Upadacitinib 15 mg QD and subjects switching from methotrexate (MTX) to Upadacitinib 15 mg QD.

#### 3. Upadacitinib 30 mg QD

This includes Upadacitinib 30 mg QD exposure from subjects starting on Upadacitinib 30 mg QD and subjects switching from MTX to Upadacitinib 30 mg QD. Exposure is censored at time of dose switch from Upadacitinib 30 mg QD to Upadacitinib 15 mg QD.

4. Upadacitinib 15 mg QD switched from Upadacitinib 30 mg QD

This includes Upadacitinib 15 mg QD exposure from subjects who switched dose from Upadacitinib 30 mg QD to Upadacitinib 15 mg QD.

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD. Exposure to upadacitinib 30 mg QD (Group 3) will be censored prior to the day subject received the first dose of upadacitinib 15 mg QD, and subsequent exposure to upadacitinib 15 mg QD will be summarized under a separate group (Group 4).

The duration of exposure to study drug will be summarized for each group as specified above, with the number of subjects, mean, standard deviation, median, minimum and maximum values. In addition, the number and percentage of subjects exposed to study drug will be summarized for the following cumulative duration intervals.

- $\geq 2$  weeks
- $\geq$  4 weeks
- > 14 weeks
- $\geq$  26 weeks
- $\geq$  36 weeks

- > 52 weeks
- $\geq 78$  weeks
- $\geq 2$  years
- $\geq 2.5$  years
- $\geq 3$  years
- $\geq$  4 years

### 7.2 Compliance

Study drug compliance for Upadacitinib/PBO and for MTX/PBO will be summarized separately for each treatment group for Period 1. Upadacitinib/PBO compliance is defined as the number of Upadacitinib/PBO tablets taken (i.e., the difference between the number of tablets dispensed and the number of tablets returned) during the subject's participation in Period 1 divided by the number of days that the subject was in the Treatment Phase of Period 1. MTX/PBO compliance is defined as the number of MTX doses taken during the subject's participation in Period 1 divided by the number of weeks that the subject was in the Treatment Phase of Period 1.

# 8.0 Efficacy Analysis

#### 8.1 General Considerations

There are two sets of planned efficacy analysis: efficacy analysis for Period 1 and long-term efficacy analysis. All efficacy analyses will be carried out using the FAS population.

## 8.1.1 Efficacy Analysis at Different Phases of the Study

#### **Efficacy Analysis for Period 1**

Standard efficacy analysis by randomized treatment groups (Upadacitinib 15 mg QD, Upadacitinib 30 mg QD and the combined MTX groups) will be performed on efficacy data up to Week 14. No protocol-defined treatment switching will occur prior to the time



point. Formal statistical inference will be generated, and results from this set of analysis will be used as the key efficacy findings of this study.

#### **Long-Term Efficacy Analysis**

Long-term efficacy analysis will be performed on As Observed data (defined in Section 8.1.2) by randomized treatment group sequence as described below:

- 1.  $MTX \rightarrow Upadacitinib 15 mg QD$
- 2. MTX → Upadacitinib 30 mg QD
- 3. Upadacitinib 15 mg QD
- 4. Upadacitinib 30 mg QD

There will be no statistical testing; only descriptive statistics and confidence intervals will be provided.

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD. For long-term efficacy analysis, subjects will continue to be summarized under the treatment sequences as described above, regardless of dose switch – i.e., for treatment sequences 2 and 4, data collected after dose switch will continue to be summarized under the same treatment sequences. The visit at which dose switch occurs could be different for each subject. The first and last visits at which dose switch occurs will be noted in the summary.

#### 8.1.2 Definition of Missing Data Imputation

#### Non-Responder Imputation (NRI) Approach

The NRI approach will categorize any subject who has missing value for categorical variables at a specific visit as non-responder for that visit. In addition, subjects who prematurely discontinue from study drug will be considered as non-responders for all subsequent visits after discontinuation.



#### **Observed Cases (OC)**

The OC analysis will not impute values for missing evaluations. In addition, the OC will not use values after premature discontinuation of study drug. This sensitivity analysis will only be applied to the analysis prior to treatment switching.

#### As Observed (AO)

The AO analysis will not impute values for missing evaluations. Regardless of treatment switching or premature discontinuation of study drug, all observed data will be used in the analysis. The AO analysis will be applied to long-term efficacy analysis.

#### Mixed Effect Model Repeat Measurement (MMRM) for Short-Term Analysis

The repeated measure analysis will be conducted using mixed model including observed measurements at all visits. The mixed model includes the categorical fixed effects of treatment, visit and treatment-by-visit interaction, main stratification factors at randomization and the continuous fixed covariates of baseline measurement. An unstructured variance covariance matrix will be used. The parameter estimations are based on the assumption of data being missing at random and using the method of restrictive maximum likelihood (REML). The missing at random assumption is considered reasonable given the high placebo response rate typically seen in RA trials. Additionally in RA trials, the proportion of discontinuation is relatively small (10 - 15%) only) and the rate of discontinuation due to lack of efficacy is generally low (< 5%).

#### MMRM and Generalized Linear Mixed Model (GLMM) for Long-Term Analysis

The repeated measure analysis will be conducted using mixed model including As Observed measurements at all visits. MMRM will be used for continuous endpoints and GLMM will be used for binary endpoints. The mixed models will include the categorical fixed effects of treatment, visit and treatment-by-visit interaction, and main stratification factor geographic region. For the MMRM analysis of change from baseline in continuous endpoints, the baseline measurement will be included as a continuous fixed covariate. The categorical fixed effect of subject's discontinuation status may also be included in the



model as appropriate. Unstructured, Toeplitz, compound symmetry, or other covariance structures may be considered.

#### **Multiple Imputation (MI)**

The MI analysis will impute missing data multiple times under appropriate random variation and thus generate multiple imputed "pseudo-complete" datasets. Results will be aggregated across the multiple imputed datasets, overcoming drawbacks of the single imputation methods. LOCF will be first applied to augment data into monotonic missing pattern and PROC MI will be used to generate 5 datasets using the regression method. Specifically, visits will be imputed in order, where later visits are imputed by regressing upon all previous visits, baseline, treatment group, demographics and other key baseline characteristics. Analysis will first be performed on each of the multiple imputed datasets, and PROC MIANALYZE will then be used to aggregate the results for the final statistical inference. The imputation is based on assumption of data being missing at random. The missing at random assumption is considered reasonable given the high placebo response rate typically seen in RA trials. Additionally in RA trials, the proportion of discontinuation is relatively small (10 – 15% only) and the rate of discontinuation due to lack of efficacy is generally low (< 5%).

The NRI approach will serve as the primary analysis approach for key binary endpoints while OC will also be repeated as a sensitivity analysis. The MI approach will serve as the primary analysis approach for key continuous endpoints HAQ-DI and DAS28. The MMRM will serve as the primary analysis for other key continuous endpoints. A missing not at random (MNAR) model that varies assumptions for the missing data in active treatment groups and placebo groups may be used as a sensitivity analysis for key continuous endpoints at Week 14 to account for potential deviation from the MAR assumption. The AO analysis will be performed for descriptive summary.



#### 8.2 Efficacy Analysis for Period 1

#### 8.2.1 Primary Efficacy Analysis

The primary endpoint for US/FDA regulatory purposes is ACR20 response at Week 14. The primary endpoint for EU/EMA regulatory purposes is LDA (based on DAS28 (CRP) ≤ 3.2) at Week 14. Analyses will be conducted separately for US/FDA regulatory purposes and EU/EMA regulatory purposes; for each set of analysis, only one primary endpoint is specified.

Analysis of the primary endpoint will be conducted on the FAS based on randomized treatment groups (Upadacitinib 15 mg QD, Upadacitinib 30 mg QD and the combined MTX groups). Point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Comparisons of the primary endpoint will be made between each Upadacitinib dose and the combined MTX group using the Cochran-Mantel-Haenszel test adjusting for stratification factor geographic region. Point estimate, 95% CI using normal approximation and p-value for the treatment comparison will be presented. Both nominal p-value constructed using the Cochran-Mantel-Haenszel test and adjusted p-value through the graphical multiplicity procedure described in Section 8.2.5 will be provided. For the primary analysis, non-responder imputation (NRI) will be used.

# 8.2.2 Sensitivity Analysis of Primary Efficacy Variables

The primary analysis for point estimate and CI will be repeated using Observed Cases without any imputation as a sensitivity analysis. This will be conducted on the FAS based on randomized treatment groups.

Supportive NRI analysis will also be conducted on the Per Protocol Analysis Set.

### 8.2.3 Key Secondary Efficacy Analyses

Ranked key secondary endpoints (at Week 14) for US/FDA regulatory purposes are:



- 1. Change from baseline in DAS28 (CRP);
- 2. Change from baseline in HAQ-DI;
- 3. Change from baseline in SF-36 Physical Component Score (PCS);
- 4. Proportion of subjects achieving LDA based on DAS28 (CRP)  $\leq$  3.2;
- 5. Proportion of subjects achieving Clinical remission (CR) based on DAS28 (CRP);
- 6. Change from baseline in morning stiffness (duration).

Ranked key secondary endpoints (at Week 14) for EU/EMA regulatory purposes are:

- 1. Change from baseline in DAS28 (CRP);
- 2. Change from baseline in HAQ-DI;
- 3. ACR20 response rate;
- 4. Change from baseline in SF-36 PCS;
- 5. Proportion of subjects achieving CR based on DAS28 (CRP);
- 6. Change from baseline in morning stiffness (duration).

Other key secondary endpoints (at Week 14) for both US/FDA and EU/EMA regulatory purposes are:

- 1. ACR50 response rate;
- 2. ACR70 response rate;

For binary endpoints, frequencies and percentages will be reported for each randomized treatment group. Similar analyses as for the primary endpoint will be conducted.

For the major RA continuous endpoints DAS28 and HAQ-DI change from baseline, statistical inference will be conducted using analysis of covariance (ANCOVA) coupled with MI for missing data handling. Specifically, the ANCOVA model will include

treatment as the fixed factor, and the corresponding baseline value and the stratification factor geographic region as the covariates. For other continuous endpoints, statistical inference will be conducted using the MMRM model as described in Section 8.1.2, with the main stratification factor being geographic region. From both the MI and MMRM analyses, the LS mean and 95% CI will be reported for each randomized treatment group; the LS mean treatment difference and associated 95% CI and p-value will be reported comparing each Upadacitinib dose group with the combined MTX group. Both nominal p-value and adjusted p-value through the graphical multiplicity procedure described in Section 8.2.5 will be provided.

#### 8.2.4 Exploratory Efficacy Analyses

Additional efficacy analysis includes the following endpoints at Week 2, 4, 8, and 14 are:

- Change from baseline in individual components of ACR response;
- ACR20/50/70 response rates;
- Change from baseline in DAS28 (CRP) and DAS28 (erythrocyte sedimentation rate [ESR]);
- Change from baseline in CDAI and SDAI;
- Change from baseline in morning stiffness (severity and duration);
- Proportion of subjects achieving LDA and proportion of subjects achieving CR based on DAS28 (CRP), DAS28 (ESR), Simplified Disease Activity Index (SDAI), and CDAI criteria (see below);
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.3 among those with baseline HAQ-DI  $\geq$  0.3;
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.22 among those with baseline HAQ-DI  $\geq$  0.22;
- ACR/EULAR Boolean remission;

| | DAS28 (CRP) and DAS28 (ESR) | SDAI | CDAI |
|-----|-----------------------------|--------|-------|
| LDA | ≤ 3.2 | ≤ 11.0 | ≤ 10 |
| CR | < 2.6 | ≤ 3.3 | ≤ 2.8 |



Additional endpoints at Weeks 4 and 14 are:

- Change from baseline in EQ-5D-5L;
- Change from baseline in SF-36.

For binary endpoints, point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Point estimate, 95% CI and p-value will be provided for the treatment comparison between each Upadacitinib dose group and the combined MTX group using the Cochran-Mantel-Haenszel test adjusting for stratification factor geographic region. Only the nominal p-value will be provided, and the 95% CI will be based on normal approximation. NRI will be used as primary analysis and OC will be used as sensitivity analysis.

For continuous endpoints, the LS mean and 95% CI will be reported for each randomized treatment group. The LS mean treatment difference and associated 95% CI and p-values between each Upadacitinib dose group and the combined MTX group will be provided using MMRM model with fixed effects of treatment, visit and treatment-by-visit interaction, geographic region and baseline value as covariate. Only the nominal p-value will be provided.

#### 8.2.5 Handling of Multiplicity

The overall type I error rate of the primary and ranked key secondary endpoints for the two doses will be strongly controlled using a graphical multiple testing procedure. Specifically, the testing will utilize the endpoint sequence of primary endpoint followed by the ranked key secondary endpoints in the order as specified in Section 8.2.3, and will begin with testing the primary endpoint using  $\alpha$  of 0.025 for each dose. Continued testing will follow a pre-specified  $\alpha$  transfer path which includes downstream transfer along the endpoint sequence within each dose as well as cross-dose transfer. Adjusted p-values for the primary and ranked key secondary endpoints will be provided based on the testing procedure.



The graphs for the testing procedures are provided in Figure 3 and Figure 4, for US/FDA and EU/EMA regulatory purposes, respectively. In the graph, the arrows specify the  $\alpha$  transfer paths. Once an endpoint is rejected (i.e., deemed significant) at its assigned significance level, its significance level will be transferred to subsequent endpoint(s) following the arrow(s). If more than one arrow originates from an endpoint, the significance level for this endpoint (once rejected) will be split between multiple subsequent endpoints following the arrows. The numbers on the arrows denote the weights for transferring and (possibly) splitting significance levels. Specifically, the weight 1 denotes 100% transfer of significance level, and the weight  $\frac{1}{2}$  denotes 50 – 50% splitting of significance level.

Figure 3. Graphical Multiple Testing Procedure for US/FDA Regulatory Purposes



Figure 4. Graphical Multiple Testing Procedure for EU/EMA Regulatory Purposes



# 8.2.6 Efficacy Subgroup Analysis

The primary efficacy endpoint will be examined in the subgroups listed in Table 4 below. Treatment difference between each Upadacitinib dose and the combined MTX group will be presented with point estimate and 95% confidence interval using normal approximation. No p-value will be provided for subgroup analysis. If any of the resulting


subgroups has fewer than 10% of the planned study size (i.e., < 60 subjects), the subgroup analyses for that variable will not be presented.

Table 4. Subgroups for Efficacy Analysis

| Subgroup Factor | Categories |
|---|---|
| Age | < 40, [40, 65], ≥ 65 |
| Sex | Male or Female |
| Weight | $< 60 \text{ kg or} \ge 60 \text{ kg}$ |
| BMI | $< 25 \text{ or } \ge 25$ |
| Race | White, Black or African American, American Indian or Alaska<br>Native, Native Hawaiian or Other Pacific Islander, Asian, Other |
| Geographic Region | North America, South/Central America, Western Europe, Eastern Europe, Japan, Other |
| Duration of RA disease diagnosis | $< 5$ year or $\ge 5$ year |
| Baseline Rheumatoid Factor<br>Status | Positive or Negative |
| Baseline Anti-CCP Antibody<br>Status | Positive or Negative |
| Baseline RF and Anti-CCP | At least one positive or double negative |
| Baseline DAS28 [hsCRP] | $\leq 5.1 \text{ or} > 5.1$ |

# 8.2.7 Summary of Efficacy Analysis for Period 1

Table 5 below provides the overview of the efficacy analyses in Period 1 to be performed on different endpoints.



# Table 5. Summary of Efficacy Variables and Corresponding Analyses for Efficacy Analysis in Period 1

| Efficacy Variables | Analysis Method |
|---|---|
| Primary Variables | |
| <ul> <li>ACR20 response at Wee</li> <li>LDA as measured by DA at Week 14<sup>b</sup></li> </ul> | |
| | group, where the p-value is constructed using the Cochran-Mantel-Haenszel test adjusting for stratification factor geographic region. Both nominal p-value and adjusted p-value through the graphical multiplicity procedure described in Section 8.2.5 will be provided. The 95% CI will be based on normal approximation. |
| | <ul> <li>Subgroup analysis.</li> <li>Imputation: NRI for primary analysis and OC for sensitivity analysis</li> </ul> |
| | <ul> <li>Analysis Set: FAS and Per Protocol Analysis Set as supportive<br/>analysis (NRI only).</li> </ul> |
| Key Secondary Variables | |
| Binary Endpoints: • ACR50/70 response at V | • Point estimate and 95% CI of the response rate for each treatment group. The 95% CI will be based on normal approximation. |
| <ul> <li>ACR 20 response at Wee</li> <li>CR as measure by DAS2<br/>Week 14</li> </ul> | • Point estimate, 95% CI and p-value for the treatment comparison between each Upadacitinib dose group and the combined MTX group using the Cochran-Mantel-Haenszel test adjusting for |
| • LDA as measured by DA at Week 14 <sup>a</sup> | AS28 (CRP) stratification factor geographic region. For ranked key secondary endpoints, both nominal p-value and adjusted p-value through the graphical multiplicity procedure described in Section 8.2.5 will be provided. The 95% CI will be based on normal approximation. |
| | <ul> <li>Imputation: NRI for primary analysis and OC for sensitivity analysis</li> </ul> |
| | Analysis Set: FAS |
| <ul> <li>Continuous Endpoints:</li> <li>Change from baseline in DAS28(CRP) at Week 1</li> <li>Change from baseline in Week 14</li> </ul> | 4 combined MTX group using ANCOVA model with treatment, |



# Table 5. Summary of Efficacy Variables and Corresponding Analyses for Efficacy Analysis in Period 1 (Continued)

| Efficacy Variables | Analysis Method |
|---|---|
| Key Secondary Variables (continued) | |
| <ul> <li>Change from baseline in SF-36 Physical Component Score (PCS) at Week 14 </li> <li>Change from baseline in morning stiffness (duration) at Week 14</li> </ul> | <ul> <li>LS mean and 95% CI within each treatment group and LS mean, 95% CI and p-values between each Upadacitinib dose group and the combined MTX group using MMRM model with fixed effects of treatment, visit and treatment-by-visit interaction, geographic region and baseline value as covariate. Both nominal p-value and adjusted p-value through the graphical multiplicity procedure described in Section 8.2.5 will be provided.</li> <li>Analysis Set: FAS</li> </ul> |
| Additional Variables (Summarized at Al | Visits Up to Week 14) |
| <ul> <li>Binary Endpoints:</li> <li>ACR20/50/70 response</li> <li>LDA and CR based on DAS28 (CRP), DAS28 (ESR), SDAI, and CDAI criteria</li> <li>Proportion of subjects with change from baseline in HAQ-DI ≤ -0.3 among those with baseline HAQ-DI ≥ 0.3;</li> <li>Proportion of subjects with change from baseline in HAQ-DI ≤ -0.22 among those with baseline HAQ-DI ≥ 0.22;</li> <li>ACR/EULAR Boolean remission</li> </ul> | <ul> <li>Point estimate and 95% CI of the response rate for each treatment group. The 95% CI will be based on normal approximation.</li> <li>Point estimate, 95% CI and p-value for the treatment comparison between each Upadacitinib dose group and the combined MTX group using the Cochran-Mantel-Haenszel test adjusting for stratification factor geographic region. Only nominal p-value will be provided, and the 95% CI will be based on normal approximation.</li> <li>Imputation: NRI for primary analysis and OC for sensitivity analysis</li> <li>Analysis Set: FAS</li> </ul> |
| <ul> <li>Continuous Endpoints:</li> <li>Change from baseline in individual ACR components</li> <li>Change from baseline in DAS28 (CRP) and DAS28 (ESR)</li> <li>Change from baseline in CDAI and SDAI</li> <li>Change from baseline in morning stiffness (severity and duration)</li> <li>Change from baseline in EQ-5D-5L</li> <li>Change from baseline in SF-36</li> </ul> | <ul> <li>LS mean and 95% CI within each treatment group and LS mean, 95% CI and p-values between each Upadacitinib dose group and the combined MTX group using MMRM model with fixed effects of treatment, visit and treatment-by-visit interaction, geographic region and baseline value as covariate. Only nominal p-value will be provided.</li> <li>Analysis Set: FAS</li> </ul> |

- $a. \hspace{0.5cm} US/FDA \hspace{0.1cm} regulatory \hspace{0.1cm} purposes.$
- b. EU/EMA regulatory purposes.



# 8.3 Long-Term Efficacy Analyses

Assessments to evaluate long-term efficacy will be analyzed for the following measures at Week 2, 4, 8, 14, 20, 26, 36, 48, every 12 weeks through Week 240, and at Week 260.

- ACR20/50/70 response rates;
- Change from baseline in individual ACR components;
- Change from baseline in DAS28 (CRP);
- Change from baseline in DAS28 (ESR);
- Change from baseline in CDAI;
- Change from baseline in SDAI;
- Change from baseline in morning stiffness (severity and duration);
- Proportion of subjects achieving LDA and proportion of subjects achieving CR based on DAS28 (CRP), DAS28 (ESR), SDAI, and CDAI criteria;
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.3 among those with baseline HAQ-DI  $\geq$  0.3;
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.22 among those with baseline HAQ-DI  $\geq$  0.22;
- ACR/EULAR Boolean remission;
- Proportion of subjects with no concomitant corticosteroid use (among subjects with corticosteroid use at baseline).

Assessments to evaluate long-term efficacy will be analyzed for the following measures at Week 4, 14 and 48:

- Change from baseline in EQ-5D-5L;
- Change from baseline in SF-36.

Analyses will be based on As Observed (AO) data. Descriptive statistics will be provided for each randomized treatment group sequence as defined in Section 8.1.1. These include the number of observations, mean, standard deviation, and 95% CI for continuous endpoints and frequencies and percentages with 95% CI using normal approximation for



binary endpoints. In addition, longitudinal analysis will be performed using MMRM or GLMM as described in Section 8.2.1 for all endpoints except proportion of subjects with no concomitant corticosteroid use. Point estimates and 95% CI from the model will be provided for each treatment group sequence. Plot for each randomized treatment group sequence over time will be provided.

Table 6 below provides the overview of the long-term efficacy analyses to be performed on different endpoints.



# Table 6. Summary of Efficacy Variables and Corresponding Analyses for Long-Term Efficacy Analysis

| Efficacy Variables | <b>Analysis Method</b> |
|---|---|
| Binary Endpoints: | |
| <ul> <li>ACR20/50/70 response by visit</li> <li>LDA and CR based on DAS28 (CRP),<br/>DAS28 (ESR), SDAI, and CDAI criteria<br/>by visit</li> <li>Proportion of subjects with change from<br/>baseline in HAQ-DI ≤ -0.3 and ≤ -0.22,<br/>respectively</li> <li>ACR/EULAR Boolean remission by visit</li> <li>Proportion of subjects with no concomitant<br/>corticosteroid use (among subjects with<br/>corticosteroid use at baseline)*</li> </ul> | <ul> <li>Point estimate and 95% CI of the response rate for each randomized treatment group sequence</li> <li>Point estimate and 95% CI of the response rate using GLMM model for each randomized treatment group sequence (*endpoint excluded from this analysis)</li> <li>Plot for each randomized treatment group sequence over time for key endpoints#</li> <li>Imputation: AO</li> <li>Analysis Set: FAS</li> </ul> |
| <b>Continuous Endpoints:</b> | |
| <ul> <li>Change from baseline in individual ACR components by visit</li> <li>Change from baseline in DAS28 (CRP) and DAS28 (ESR) by visit</li> <li>Change from baseline in CDAI and SDAI by visit</li> <li>Proportion of subjects with change from baseline in HAQ-DI ≤ -0.3 by visit</li> <li>Proportion of subjects with change from baseline in HAQ-DI ≤ -0.22 by visit</li> <li>Change from baseline in morning stiffness (severity and duration) by visit</li> <li>Change from baseline in EQ-5D-5L by visit</li> </ul> | <ul> <li>Point estimate, and 95% CI of mean change from baseline together with SD for each randomized treatment group sequence</li> <li>Point estimate and 95% CI of change from baseline using MMRM model for each randomized treatment group sequence</li> <li>Plot for each randomized treatment group sequence over time for key endpoints#</li> <li>Imputation: AO</li> <li>Analysis Set: FAS</li> </ul> |
| <ul> <li>Change from baseline in SF-36 by visit</li> </ul> | |

Key endpoints for figures include: ACR20/50/70, LDA and CR based on DAS28(CRP) and CDAI criteria, Boolean remission, change from baseline in DAS28(CRP) and CDAI.

# 8.4 Efficacy Variables Definitions and Conventions

### 8.4.1 ACR Criteria

ACR criteria are a commonly used standard criteria set mentioned in the guidance of American College of Rheumatology to evaluate the effectiveness of investigation drug in



RA clinical trials. It is a composite measurement calculated based on the improvement over a set of core measurements.

ACR20 is defined as at least 20% improvement (compared to baseline values) in tender and swollen joint counts and at least 20% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function and acute phase reactant hsCRP).

ACR50 and ACR70 are similarly defined with at least 50% and 70% improvement, respectively.

A subject will be classified as an ACR20 (ACR50, ACR70) responder, if the following conditions are met:

- 1.  $\geq$  20% (50%, 70%) improvement from baseline in tender joint count (TJC68) and
- 2.  $\geq 20\%$  (50%, 70%) improvement from baseline in swollen joint count (SJC66) and
- 3.  $\geq 20\%$  (50%, 70%) improvement from baseline in at least 3 of the following 5:
  - patient's assessment of pain
  - patient's global assessment of disease activity (PGA)
  - physician's global assessment of disease activity (PhGA)
  - patient's self-assessment of physical function (i.e., measured by Health Assessment Questionnaire (HAQ-DI score)
  - Acute-phase reactant value CRP

There are seven components to be evaluated to define an ACR response. Missing values for each component can occur due to a missed visit or due to dropout from the study. Depending on the pattern of the missing components, ACR responses may be or may not be determined using observed values only.

To maximize the utilization of observed information at certain visits and be scientifically as robust as possible, the principle to calculate ACR response is to minimize imputation whenever possible. Observed ACR response will be calculated first based on a derived visit window instead of the nominal visit identifier (e.g., Week 6 visit) collected from the CRF.

### To calculate observed ACR responses:

- Identify the observed component xx% improvement indicator (0/1/missing), 1 means achieving  $\ge xx\%$  improvement from baseline and 0 means < xx% improvement from baseline (e.g., xx% representing 20%/50%/70%).
- ACRxx = 0 if TJC indicator = 0 OR SJC indicator = 0 OR at least 3 out of 5 components improvement indicators = 0.
- ACRxx = 1 if TJC indicator = 1 AND SJC indicator = 1 AND at least 3 out of 5 components improvement indicators = 1.
- For all other cases, ACRxx = missing since ACRxx cannot be determined.

The following table illustrates examples for ACR calculations.

| Example | TJC<br>68 | SJC<br>66 | Component 1 | Component 2 | Component 3 | Component 4 | Component 5 | ACR20-<br>Response? |
|---|---|---|---|---|---|---|---|---|
| A | 1 | 1 | 1 | 1 | 1 | | | Yes |
| В | 1 | 0 | 1 | 1 | 1 | 1 | 1 | No |
| C | | 0 | | | | | | No |
| D | 1 | | 1 | 1 | 1 | 1 | 1 | |
| E | 1 | 1 | 0 | 0 | 0 | 1 | 1 | No |
| F | | | 0 | 0 | 0 | | | No |
| G | 1 | 1 | 1 | 1 | 0 | 0 | • | |

Legend: 1 = 20% improved compared to baseline; 0 = 20% improved compared to baseline; "." missing

### Windowing Rule for ACR Response Calculation:

• ACR component values will first be determined at each date within a visit window.



- ACR component values at each date will be combined to determine the observed ACR composite score at each date in each window.
- After this calculation, if multiple non-missing ACR composite scores are
  available within a given visit window, the non-missing ACR composite score
  closest to the target day will be used. If two composite scores have the same
  distance from the target day, the later one will be used. The corresponding
  date will be used as the observed ACR response date in the derived efficacy
  dataset.
- If a non-missing ACR composite score is not available for any day within a given visit window, the windowed component values for that visit will be used to calculate the ACR composite score for that visit window (component value windowing follow the same rules as in steps described above). The date of observed ACR composite score will be determined by the first available ACR component date, in the order of TJC, SJC, Pain, PGA, PhGA, HAQ-DI, CRP/ESR, in the derived efficacy dataset.

When observed ACR xx response for a given visit is missing, imputation methods will be used to calculate "imputed" ACRxx response.

Non-Responder Imputation (NRI) for ACR response:

- Step 1: all missing components will be imputed using LOCF, and then the ACR composite score can be calculated.
- Step 2: if the ACR composite score cannot be determined by step 1, the ACR composite score will be imputed as 0. In addition, subjects who prematurely discontinue from the study drug will be considered as nonresponders (ACR = 0) for all subsequent visits after the discontinuation date.

#### 8.4.2 Joint Evaluation

Anatomical joints are evaluated for swelling and tenderness at every study visit. The 34 anatomical joints in Table 7 are assessed in this study for both the left and right side of the body.



Table 7. Anatomical Joints Assessed for Calculation of Tender and Swollen Joint Counts (TJC68 and SJC66)

| Temporomandibular | Sternoclavicular | Acromio-clavicular | Shoulder |
|---|---|---|---|
| Elbow | Wrist | Metacarpophalangeal I | Metacarpophalangeal II |
| Metacarpophalangeal<br>III | Metacarpophalangeal IV | Metacarpophalangeal V | Thumb Interphalangeal |
| Proximal<br>Interphalangeal II | Proximal<br>Interphalangeal III | Proximal<br>Interphalangeal IV | Proximal<br>Interphalangeal V |
| Distal Interphalangeal II | Distal<br>Interphalangeal III | Distal<br>Interphalangeal IV | Distal<br>Interphalangeal V |
| Hip <sup>a</sup> | Knee | Ankle | Tarsus |
| Metatarsophalangeal I | Metatarsophalangeal<br>II | Metatarsophalangeal III | Metatarsophalangeal IV |
| Metatarsophalangeal V | Great Toe/Hallux | Interphalangeal II | Interphalangeal III |
| Interphalangeal IV | Interphalangeal V | | |

a. Hip joints are not assessed for swelling.

At each study visit, a joint evaluator assessed whether a particular joint was "tender or painful" where presence of tenderness was scored as "1" and the absence of tenderness was scored as "0," provided the joint was not replaced ("9") or could not be assessed ("NA") due to other reasons (e.g., post-corticosteroid joint injection). The total tender joint count (TJC68), which is based on 68 joints, will be derived as the sum of all "1s" and proportional extrapolation will be used to impute joint counts for the joints that are replaced or not assessed. A similar method will be followed for the derivation of total swollen joint count (SJC66), which is based on 66 joints as the hip joints are excluded. Thus, the range for TJC68 will be 0 to 68 and 0 to 66 for SJC66.

# 8.4.3 Patient's Global Assessment of Disease Activity Visual Analog Scale (VAS)

The subject will assess his/her disease activity for the past 24 hours using a Patient's Global Assessment of Disease VAS. The range is 0 to 100 mm with no activity being indicated by 0 and severe activity by 100.

# 8.4.4 Physician's Global Assessment of Disease Activity Visual Analog Scale (VAS)

The physician will assess Patient's disease activity at the time of visit using a Physician's Global Assessment of Disease VAS. The range is 0 to 100 mm with no activity being indicated by 0 and severe activity by 100.

### 8.4.5 Patient's Global Assessment of Pain

The subject will assess his/her pain in the previous week using a Patient's Global Assessment Pain VAS. The range is 0 to 100 mm with no pain being indicated by 0 and severe pain by 100.

# 8.4.6 Disease Activity Score (DAS28)

DAS28 (CRP) and DAS28 (ESR) are composite indices to assess disease activity in RA patients using hsCRP or ESR measurement respectively. The DAS provides a score between 0 and 10, indicating how active the rheumatoid arthritis is at the time of measurement.

DAS28 (CRP) and DAS28 (ESR) can be calculated based on Tender Joint Count, Swollen Joint Count, Patient's Global Assessment of Disease Activity (PtGA) (in mm), and hsCRP (in mg/L) or ESR (mm/hr).

DAS28 (CRP) = 
$$0.56 \times \sqrt{\text{TJC28*}} + 0.28 \times \sqrt{\text{SJC28**}} + 0.36 \times \ln(\text{hsCRP}^{\&} + 1) + 0.014 \times \text{PtGA}^{\circ} + 0.96$$

DAS28 (ESR) = 
$$0.56 \times \sqrt{\text{TJC28*}} + 0.28 \times \sqrt{\text{SJC28**}} + 0.70 \times \ln(\text{ESR}^{\#}) + 0.014 \times \text{PtGA}^{"}$$

- \* TJC28 refers to the Subject's total Tender Joint Count out of the provided 28 evaluated joints.
- \*\* SJC28 refers to the Subject's total Swollen Joint Count out of the provided 28 evaluated joints.
- & hsCRP refers to the high-sensitivity c-reactive protein lab value. hsCRP unit in the DAS28 (CRP) equation is expressed as mg/L.
- # ESR refers to the Erythrocyte sedimentation rate. ESR unit in the DAS28 (ESR) equation is expressed as mm/hr.
- » PtGA refers to the Patient's Global Assessment of Disease Activity. where √ is square root and ln is natural log.



Table 8. Anatomical Joints for DAS28 (CRP) Calculation

| Shoulder | Elbow | Wrist | Thumb Interphalangeal |
|---|---|---|---|
| Metacarpophalangeal<br>I | Metacarpophalangeal II | Metacarpophalangeal<br>III | Metacarpophalangeal IV |
| Metacarpophalangeal<br>V | Proximal<br>Interphalangeal II | Proximal<br>Interphalangeal III | Proximal Interphalangeal<br>IV |
| Proximal<br>Interphalangeal V | Knee | | |

To calculate observed DAS28 scores, the observed component value will be calculated first. Then the components will be included in the calculation per the DAS formula selected. If any observed component is missing in a window, then the observed DAS28 score will be missing.

# 8.4.7 Simplified Disease Activity Index (SDAI)

SDAI is a composite continuous index to assess disease activity based on TJC28, SJC28, Patient's Global Assessment of Disease Activity (PtGA) (in cm, 0 - 10), Physician's Global Assessment of Disease Activity (PhGA) (in cm, 0 - 10) and hsCRP (mg/dL). It can be derived as follows:

$$SDAI = TJC28 + SJC28 + PtGA (cm) + PhGA (cm) + hsCRP (mg/dL).$$

To calculate observed SDAI scores, the observed component value will be calculated first. Then the components will be included in the calculation per the SDAI formula selected. If any observed component is missing in a window, then the observed SDAI score will be missing.

### 8.4.8 Clinical Disease Activity Index (CDAI)

CDAI is a composite continuous index to assess disease activity without using hsCRP measurement. It can be calculated based on TJC28, SJC28, Patient's Global Assessment of Disease Activity (PtGA) (in cm, 0-10) and Physician's Global Assessment of Disease Activity (PhGA) (in cm, 0-10). It can be derived as follows:



$$CDAI = TJC28 + SJC28 + PtGA (cm) + PhGA (cm).$$

To calculate observed CDAI scores, the observed component value will be calculated first. Then the components will be included in the calculation per the CDAI formula selected. If any observed component is missing in a window, then the observed CDAI score will be missing.

# 8.4.9 Clinical Remission (CR) and Low Disease Activity (LDA)

Clinical remission (CR) and low disease activity (LDA) based on DAS28 (CRP), DAS28 (ESR), SDAI and CDAI are defined as follows:

| | DAS28 (CRP) and DAS28 (ESR) | SDAI | CDAI |
|-----|-----------------------------|--------|-------|
| LDA | ≤ 3.2 | ≤ 11.0 | ≤ 10 |
| CR | < 2.6 | ≤ 3.3 | ≤ 2.8 |

#### 8.4.10 ACR/EULAR Boolean Remission

ACR/EULAR Boolean remission is defined based on the following four criteria:

- Tender joint count  $\leq 1$  (based on 28 joints)
- Swollen joint count  $\leq 1$  (based on 28 joints)
- $CRP \le 1 \text{ mg/dL}$
- Patient global assessment of disease activity  $\leq 10$  (mm)

All four criteria must be satisfied at a visit for a subject to be classified as achieving ACR/EULAR Boolean remission.

# 8.4.11 Disability Index of Health Assessment Questionnaire (HAQ-DI)

HAQ-DI is a self-reported patient outcome measurement. It is calculated as the mean of the scores from 8 following categories with a range 0-3: Dressing and Grooming,



Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. The higher the score, the more likely to associate with morbidity and mortality for the RA patient.

The maximum score for all the questions in each category is considered as the score for the category. The Standard disability index (HAQ-DI) takes into account the subject's use of aids or devices or assistance in the scoring algorithm for a disability category. For each of the eight disability categories there is an AIDS OR DEVICES companion variable(s) that is used to record the type of assistance, if any, a subject uses for his/her usual activities. If aids or devices and/or assistance from another person are checked for a disability category, the score for this category is set to 2 (much difficulty), if the original score is 0 (no difficulty) or 1 (some difficulty). The HAQ-DI is then calculated by summing the adjusted categories scores and dividing by the number of categories answered. The HAQ-DI cannot be calculated if the patient does not have scores for at least 6 categories.

# 8.4.12 EuroQoL-5D (EQ-5D-5L)

EQ-5D is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D consists of 2 pages. The first page measures 5 dimensions of the health status (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with 5 levels per dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems corresponding to Level 1 to Level 5 respectively). The second page is an EQ Visual Analogue Scale (EQ VAS). EQ-5D health states, defined by the EQ-5D-5L descriptive system on the first page, may be converted into a single index value. The change from baseline of the index value and EQ VAS will be analyzed and reported. UK scoring algorithm will be used.

### 8.4.13 Form SF-36v2

The 36-Item Short Form, Version 2 (SF-36v2) Questionnaire with 4 week recall will be completed by the subject at Baseline, Weeks 4, 14 and 48 completion (or at PD). The SF-36v2 health survey consists of 36 general health questions and this study is using the



form for 4 weeks recall period (standard form). It has 2 components: physical and mental. For each component, a transformed summary score is calculated using 8 sub-domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.

The coding and scoring for the SF-36 will use the software provided by QualityMetrics.

# 9.0 Safety Analysis

### 9.1 General Considerations

Safety analyses will be carried out using the Safety Analysis Set. There are two sets of planned safety analysis: safety analysis for Period 1, and long-term safety analysis.

### **Safety Analysis for Period 1**

Standard safety analysis by the "as treated" treatment groups of Upadacitinib 15 mg QD, Upadacitinib 30 mg QD, and combined MTX groups will be performed on safety data up to Week 14. No protocol-defined treatment switching will occur prior to these time points.

The standard safety analyses will include reporting of adverse events (AEs), laboratory, and vital signs measurements. Frequency tables of subjects with treatment-emergent adverse events (TEAEs) by system organ class (SOC) and by preferred term (PT) as in the Medical Dictionary for Regulatory Activities (MedDRA) dictionary will be provided by treatment group. Mean changes from baseline in all continuous laboratory parameters and vital signs variables at each visit will be summarized by "as treated" treatment group. Frequency tables of subjects meeting criteria for potentially clinically significant vital sign values and for potentially clinically significant laboratory values will be provided by treatment group. Missing safety data will not be imputed.



#### **Long-Term Safety Analysis**

Long-term safety analyses that account for protocol-defined treatment switching include reporting of AE rate adjusted by cumulative exposure, mean change from baseline in laboratory parameters and vital sign variables, and rate of potentially clinically significant laboratory and vital signs values. The treatment-emergent adverse event (TEAE) rate per 100 patient-years of exposure will be presented by actual treatment received at the time of AE (as described in Section 0). Listing of subjects with TEAEs by SOC and PT will be provided. Mean changes from baseline in all continuous laboratory parameters and vital signs variables at each visit will be summarized by "as treated" treatment group sequences defined as follows (as described in Section 9.3.3 and Section 9.4.3). Frequency tables and listings of subjects meeting criteria for potentially clinically significant vital sign values and for potentially clinically significant laboratory values will be provided by actual treatment received at the time of event. Missing safety data will not be imputed.

"As treated" treatment group sequences:

- 1. MTX → Upadacitinib 15 mg QD
- 2. MTX  $\rightarrow$  Upadacitinib 30 mg QD
- 3. Upadacitinib 15 mg QD
- 4. Upadacitinib 30 mg QD

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD. For subjects who previously received upadacitinib 30 mg QD, adverse events and exposure to upadacitinib 30 mg QD will be censored at the time of dose switch; subsequent adverse events and exposure starting the day of first dose of upadacitinib 15 mg QD will be summarized under a separate group, as defined in Section 8.1. Assessment of potentially clinical significant laboratory and vital sign values will be based on the same treatment exposure groups as for adverse events, as described above. For summary of mean change from baseline in



laboratory values and vital signs, exposure sequences 2 and 4 (i.e., subjects who switched from upadacitinib 30 mg QD to 15 mg QD) will be censored at the time of dose switch. Mean change from baseline for laboratory values and vital signs collected after dose switch will be summarized separately by visits post switch.

### 9.2 Analysis of Adverse Events

A treatment-emergent Adverse Event (TEAE) is defined as an adverse event with an onset date that is after the first dose of study drug, and no more than 30 days of the drug after the last dose of study drug.

Events where the onset date is the same as the study drug start date are assumed to be treatment-emergent, unless the study drug start time and the adverse event start time are collected and the adverse event start time is prior to the study drug start time. If an incomplete onset date was collected for an adverse event, the event will be assumed to be treatment-emergent unless there is other evidence that confirms that the event was not treatment-emergent (e.g., the event end date was prior to the study drug start date).

Adverse event data will be presented by SOCs and PTs using MedDRA version 19.1. All adverse event tables will be sorted in alphabetical order by SOC and PT and descending percentages for each treatment group.

### 9.2.1 Analysis of Adverse Events for Period 1

### 9.2.1.1 Adverse Events Overview

The number and percentage of subjects experiencing TEAEs will be summarized by "as treated" treatment group and overall for the following AE categories.

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs reasonably possibly related to study drug



- TEAEs of special interest
- TEAEs leading to discontinuation of study drug
- TEAE leading to death

In the AE overview summary, any event with an unknown severity will be considered as severe and any AE with an unknown relationship will be considered as having "reasonable possibility" of being related to study drug.

Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

For TEAEs of special interest, the point estimate and 95% CI (using normal approximation) will be provided for the treatment difference in AE percentage between each Upadacitinib dose group and the combined MTX group.

As a sensitivity analysis, the AE overview summary will be repeated by randomized treatment groups. In this summary, all AEs with an onset date after the first dose of study drug will be included, regardless of whether the AE occurred more than 30 days after the last dose of study drug.

# 9.2.1.2 Adverse Events by System Organ Class and Preferred Term

The number and percentage of subjects experiencing adverse events a will be tabulated by SOC and MedDRA PT by "as treated" treatment group and overall. The SOCs will be presented in alphabetical order, and the PTs will be presented in alphabetical order within each SOC.

The following summaries of adverse events will be generated:

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs reasonably possibly related to study drug



- TEAEs leading to discontinuation of study drug
- TEAE leading to death
- Frequent AEs (reported in 2% of subjects or more in any treatment group)

Subjects reporting more than one adverse event for a given MedDRA preferred term will be counted only once for that term (most severe incident for the severity tables and most related incident for the relationship tables). Subjects reporting more than one type of adverse event within a SOC will be counted only once for that SOC. Subjects reporting more than one type of adverse event will be counted only once in the overall total.

As a sensitivity analysis, the AE summary by SOC and PT will be repeated by randomized treatment groups. In this summary, all AEs with an onset date after the first dose of study drug will be included, regardless of whether the AE occurred more than 30 days after the last dose of study drug.

### 9.2.1.3 TEAEs by Maximum Severity

TEAEs will also be summarized by maximum severity by "as treated" treatment group and overall. If a subject has an AE with an unknown severity, then the subject will be counted in the severity category of unknown, even if the subject has another occurrence of the same event with a severity present. The only exception is that if the subject has another occurrence of the same AE with the most extreme severity – severe. In this case, the subject will be counted under the severe category.

### 9.2.1.4 TEAEs by Relationship

TEAEs will also be summarized by relationship to Upadacitinib and MTX, as assessed by the investigator, by "as treated" treatment group and overall. If a subject has a TEAE with an unknown relationship, then the subject will be counted in the relationship category of "unknown," even if the subject has another occurrence of the same event with a relationship present. The only exception is if the subject has another occurrence of the same TEAE with a relationship assessment of "reasonable possibility." In this case, the subject will be counted under the "reasonable possibility" category.



# 9.2.1.5 Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term

TEAEs and reasonably possibly related AEs occurring for more than 2% of the subjects in any of the "as treated" treatment groups will be summarized by MedDRA PT in decreasing frequency separately.

# 9.2.1.6 Adverse Events of Special Interest

The Adverse Events of Special Interest (AESI) categories will be summarized and presented by "as treated" treatment group and overall using SOC and MedDRA PT. The AESI categories will be identified by the following search criteria per Standard MedDRA Queries (SMQs)/Company MedDRA Queries (CMQs) in

Table 9. AESI for Upadacitinib with SMQs/CMQs/PTs Searches

| AESI | Type of<br>MedDRA<br>Query | Broad or<br>Narrow<br>Search | SMQ/CMQ Search Criteria |
|---|---|---|---|
| Serious Infections | CMQ | | "Infections" – Subset for SAEs |
| Opportunistic Infection<br>excluding Tuberculosis and<br>Herpes Zoster | CMQ | | "Opportunistic Infection excluding<br>Tuberculosis and Herpes Zoster" |
| Possible Malignancy | SMQ | Narrow | "Malignancies" |
| Malignancy | SMQ | | "Malignant tumours" |
| Non-Melanoma Skin Cancer (NMSC) | SMQ | Narrow | Skin Malignant tumours (Narrow SMQ) removing Melanoma CMQ |
| Malignancy excluding NMSC | | | "Malignant tumours" SMQ removing NMSC output |
| Lymphoma | SMQ | | "Malignant Lymphomas" |
| Hepatic Disorder | SMQ | Narrow | "Drug Related Hepatic Disorders" |
| Adjudicated Gastrointestinal<br>Perforations | Output from adjudication | | |
| Anemia | CMQ | | "Non-Hemolytic and Non-Aplastic<br>Anemias" |
| Neutropenia | CMQ | | "Hematological Toxicity – Neutropenia" |



**Table 9.** AESI for Upadacitinib with SMQs/CMQs/PTs Searches (Continued)

| AESI | Type of<br>MedDRA<br>Query | Broad or<br>Narrow<br>Search | SMQ/CMQ Search Criteria |
|---|---|---|---|
| Lymphopenia | CMQ | | "Hematological Toxicity - Lymphopenia" |
| Herpes Zoster | CMQ | | "Herpes Zoster" |
| Creatine Phosphokinase (CPK)<br>Elevation | PT | | Search only for the PT of "Blood creatine phosphokinase increased" |
| Renal Dysfunction | SMQ | Narrow | "Acute Renal, Failure" |
| Active Tuberculosis | CMQ | | "Active Tuberculosis" |
| Adjudicated Cardiovascular<br>Events | Output from CAC | | |
| MACE* | | | |
| Cardiovascular Death | | | |
| Non-fatal Myocardial<br>Infarction | | | |
| Non-fatal Stroke | | | |
| Undetermined/Unknown<br>Cause of Deaths | | | |
| Other Cardiovascular events | | | |
| Adjudicated Thrombotic<br>Events | Output From CAC | | |
| Venous Thromboembolic<br>Events** | | | |
| Deep Vein Thrombosis | | | |
| Pulmonary Embolism | | | |
| Other Venous Thrombosis | | | |
| Arterial Thromboembolic<br>Events (non-cardiac, non-<br>neurologic) | | | |

 $CAC = Cardiovascular \ Adjudication \ Committee; \ CMQ = company \ MedDRA \ query; \ PT = preferred \ term; \ SMQ = standard \ MedDRA \ query$ 

<sup>\*</sup> MACE; Major Adverse Cardiovascular Events, defined as cardiovascular death, non-fatal myocardial infarction and non-fatal stroke.

<sup>\*\*</sup> Venous thromboembolic events (VTE) include deep vein thrombosis (DVT) and pulmonary embolism (PE) (fatal and non-fatal).



Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

# 9.2.2 Analysis of Long-Term Adverse Event Rates

Long-term adverse event rates will be analyzed using event rates adjusted by cumulative exposure and will be based on the actual treatment received at the time of AE occurrence. Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD. For subjects who previously received upadacitinib 30 mg QD, adverse events and exposure to upadacitinib 30 mg QD will be censored at the time of dose switch; subsequent adverse events and exposure starting the day of first dose of upadacitinib 15 mg QD will be summarized under a separate group. The detailed treatment groups, including the handling of dose switch, are described in Section 8.1.

# 9.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure

An overview of AEs per 100 patient-years of study exposure will be presented by treatment group and overall for the following AE categories.

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs reasonably possibly related to study drug
- TEAEs of special interest
- TEAEs leading to discontinuation of study drug
- TEAE leading to death

For this calculation, 1 year will be considered to be 365.25 days. For each treatment group, the numerator of the overall rate will be the total number of TEAEs reported for the event; that is, a subject can contribute more than one event to the numerator. For each treatment group, the denominator of the rates will be the total number of days exposed to



study drug summed across all treated subjects divided by 365.25. Please refer to Section 5.0 for the calculation of study drug exposure. The AE rate per 100 patient-years of exposure will be calculated as ([numerator/denominator])\*100. The number of AEs reported (numerator), the total number of years of study drug exposure (denominator), and the AE rate per 100 patient-years will be presented for each treatment group and overall.

Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

In the AE overview summary, any event with an unknown severity will be considered as severe and any AE with an unknown relationship will be considered as having "reasonable possibility" of being related to study drug.

For TEAEs of special interest, the point estimate and 95% CI (using normal approximation) will be provided for the treatment difference in AE rate per 100 patient-years between each Upadacitinib dose group and the combined MTX group.

# 9.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT

For each treatment group, the TEAE rate per 100 patient-years of exposure will be calculated overall, for each SOC and each PT, for each of the following events:

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs reasonably possibly related to study drug
- TEAEs leading to discontinuation of study drug
- TEAE leading to death

For this calculation, 1 year will be considered to be 365.25 days. For each treatment group, the numerator of the overall rate, the SOC rate, or the PT rate, will be the total number of TEAEs reported overall, for the SOC, or for the PT, respectively; that is a



subject can be counted more than once overall, for a SOC, and for a PT. For each treatment group, the denominator of the rates will be the total number of days exposed to study drug summed across all treated subjects divided by 365.25. Please refer to Section 5.0 for the calculation of study drug exposure. The AE rate per 100 patient-years of exposure will be calculated as [(numerator/denominator)]\*100. The number of AEs reported (numerator), the total number of years of study drug exposure (denominator), and the AE rate per 100 patient-years will be presented overall, for each SOC, and for each PT for each treatment group.

TEAE will also be summarized by MedDRA PT in decreasing frequency of the AE rate per 100 patient-years.

# 9.2.2.3 Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure

The Adverse Events of Special Interest (AESI) categories will be summarized and presented for each treatment group and overall using SOC and MedDRA PT. The AESI categories will be identified as defined in Table 9. Adjudicated cardiovascular events will be summarized and presented by treatment group using the CAC adjudicated categories.

For each treatment group, the Adverse Events of Special Interest (AESI) rate per 100 patient-years of exposure will be calculated overall, for each SOC and each PT, for each of the AESI listed in Section 9.2.1.6. For this calculation, 1 year will be considered to be 365.25 days. For each treatment group, the numerator of the overall rate, the SOC rate, or the PT rate, will be the total number of TEAEs reported overall, for the SOC, or for the PT, respectively; that is a subject can be counted more than once overall, for a SOC, and for a PT.

For each treatment group, the denominator of the rates will be the total number of days exposed to study drug summed across all treated subjects divided by 365.25. Please refer to Section 6.0 for the calculation of study drug exposure. The AE rate per 100 patient-years of exposure will be calculated as [(numerator/denominator)]\*100. The number of AEs reported (numerator), the total number of years of study drug exposure



(denominator), and the AE rate per 100 patient-years will be presented overall, for each SOC, and for each PT for each treatment group.

# 9.2.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation

All serious adverse events (SAEs), deaths, and adverse events leading to discontinuation of study drug will be listed.

# 9.3 Analysis of Laboratory Data

#### 9.3.1 Variables and Units

All laboratory parameters to be collected in this study are listed below. Laboratory parameters will be reported using the standard international (SI) units.

Table 10. List of Laboratory Variables

| <b>Laboratory Variables</b> |
|----------------------------------------------------|
| Hematology |
| White Blood Cell (WBC) Count |
| Red Blood Cell (RBC) Count |
| Hemoglobin |
| Hematocrit |
| Platelets count |
| Neutrophils |
| Basophils |
| Eosinophils |
| Lymphocytes |
| Monocytes |
| Bands |
| Chemistry |
| Total Bilirubin |
| Alkaline Phosphatase (ALP) |
| Serum glutamic oxaloacetic transaminase (SGOT/AST) |



Nitrites

# **Table 10.** List of Laboratory Variables (Continued)

| Laboratory Variables |
|--------------------------------------------------|
| Chemistry (continued) |
| Serum glutamic pyruvic transaminase (SGPT/ALT) |
| Total Protein |
| Albumin |
| Glucose |
| Triglycerides |
| Blood Urea Nitrogen (BUN) |
| Creatinine |
| Uric acid |
| Sodium |
| Potassium |
| Calcium |
| Inorganic Phosphorus |
| Creatine Phosphokinase (CPK) |
| Chloride |
| Bicarbonate |
| Cholesterol |
| LDL cholesterol |
| HDL cholesterol |
| International Normalized Ratio (INR) reflex only |
| Urinalysis |
| Specific Gravity |
| pH |
| Protein |
| Glucose |
| Ketones |
| Blood |
| Microscopic Examination (if needed) |
| Urobilinogen |
| Bilirubin |
| Leukocytes |
| 27. 1 |



### **Table 10.** List of Laboratory Variables (Continued)

| Laboratory Variables |
|----------------------------------|
| Other |
| hs-CRP |
| QuantiFERON-TB Gold <sup>a</sup> |
| IgG and IgM |
| ESR |

a. For annual follow-up QFT is captured only for those with negative QFT at Screening.

### 9.3.2 Analysis of Laboratory Data for Period 1

The laboratory data will be summarized by the "as treated" treatment groups (Upadacitinib 15 mg QD, Upadacitinib 30 mg QD, and combined MTX groups) and overall.

# 9.3.2.1 Assessment of Mean Change from Baseline and Percentage Change from Baseline in Clinical Laboratory Variables

Analyses of mean change from baseline in continuous hematology, chemistry, and urinalysis variables which are measured longitudinally will be performed by visits and by "as treated" treatment group. For each change from baseline analysis, the following summary statistics will be presented for each treatment group: sample size, baseline mean, visit mean, and the mean, standard deviation, and median of the changes from baseline. An ANOVA model with treatment as a factor will be used to test statistical significance for the change from baseline mean among different treatment groups.

In addition, similar analyses will be conducted for percentage change from baseline in LDL-C, HDL-C, TC, triglycerides, LDL-C/HDL-C ratio, TC/HDL-C ratio and hemoglobin.



# 9.3.2.2 Assessment of Shift from Baseline in Clinical Laboratory Variables

The baseline and post-baseline laboratory observations will be categorized as Grade 1, Grade 2, Grade 3, and Grade 4 according to OMERACT criteria (Rheumatology Common Toxicity Criteria v.2.0). For creatine phosphokinase and serum creatinine, NCI CTC criteria will be used.

For each laboratory variable, shift tables will be generated that cross tabulate the subjects as deemed appropriate by "as treated" treatment group:

- Category of the baseline value versus category of the final value.
- Category of the baseline value versus maximum category.
- Category of the baseline value versus minimum category.

Note that the minimum/maximum category is used, rather than the category of the minimum/maximum value. The two may be different due to variation in the reference range.

No statistical tests will be performed for this analysis.

# 9.3.2.3 Assessment of Potentially Clinical Significant Laboratory Variables

The criteria for potentially clinically significant laboratory values will be determined by OMERACT criteria of Grade 3 or 4. For creatine phosphokinase and creatinine, NCI CTC criteria will be used.

The number and percentage of subjects meeting the criteria for potentially clinically significant laboratory values will be summarized by "as treated" treatment group and overall. Only subjects with worsening in grade compare to baseline grade will be captured.



#### 9.3.2.4 Assessment of Liver Elevations

According to FDA's Guidance for Industry "Drug-Induced Liver Injury: Premarketing clinical evaluation (July 2009), when aminotransferase (AT) abnormalities indicating hepatocellular injury are accompanied by evidence of impaired hepatic function (bilirubin elevation > 2 × ULN), in the absence of evidence of biliary obstruction (i.e., significant elevation of ALP) or some other explanation of the injury (e.g., viral hepatitis, alcohol hepatitis), the combined finding (i.e., Hy's Law cases) represents a signal of a potential for the drug to cause severe DILI.

For the purpose of assessing for potential Hy's law cases, the frequencies and percentages of subjects with postbaseline liver specific function test values that meet the following criteria of potential clinical interest will be summarized by "as treated" treatment group:

- ALT  $\geq$  3 × ULN
- ALT  $\geq$  5 × ULN
- ALT  $\geq 10 \times ULN$
- ALT  $\geq 20 \times ULN$
- AST  $\geq$  3 × ULN
- AST  $\geq$  5 × ULN
- AST  $\geq 10 \times ULN$
- $AST > 20 \times ULN$
- TBL  $\geq 2 \times ULN$
- Alkaline phosphatase  $\geq 1.5 \times ULN$
- ALT and/or AST  $\geq$  3 × ULN and concurrent TBL  $\geq$  1.5 × ULN
- ALT and/or AST  $\geq 3 \times ULN$  and concurrent TBL  $\geq 2 \times ULN$



### 9.3.3 Analysis of Long-Term Laboratory Data

# 9.3.3.1 Assessment of Mean Change from Baseline and Percentage Change From Baseline in Clinical Laboratory Variables

Analyses of mean change from baseline in continuous hematology, chemistry, and urinalysis variables which are measured longitudinally will be performed by visits and by "as treated" treatment group sequences as described in Section 9.1. For each change from baseline analysis, the following summary statistics will be presented for each treatment group sequence: sample size, baseline mean, visit mean, and the mean, standard deviation, and median of the changes from baseline.

In addition, similar analyses will be performed for percentage change from baseline in LDL-C, HDL-C, triglycerides and hemoglobin.

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 QD. Mean change from baseline in laboratory values for subjects who switched from upadacitinib 30 mg QD to 15 mg QD will be censored at the time of dose switch, and mean change from baseline for values post switch will be summarized separately, as described in Section 9.1. The original study baseline will used for calculating change from baseline.

# 9.3.3.2 Assessment of Potentially Clinical Significant Laboratory Values

Long-term laboratory data will be summarized based on the number and percentage of subjects meeting the criteria for potentially clinical significant laboratory values and by the actual treatment received at the time of the event occurrence. Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 QD. The treatment groups for summarizing potentially clinical significant laboratory values are the same as the ones for long-term AE analysis as described in Section 8.1 and Section 0. A subject can be counted under different treatment groups if he/she switched treatment and experienced potentially clinical significant laboratory values under different treatment groups.



In the evaluation of potentially clinically significant laboratory values, the baseline value will be determined by the last non-missing measurement recorded on or before the date of the first dose of study drug in the corresponding treatment group (which may be different than the first dose of study drug received in the study). For example, for a subject who started on MTX and switched to Upadacitinib 15 mg QD, lab values under Upadacitinib 15 mg QD exposure would be evaluated against the baseline value defined as the last non-missing measurement recorded on or before the date of the first dose of Upadacitinib 15 mg QD. For subjects who switched from upadacitinib 30 mg QD to upadacitinib 15 mg QD, lab values under upadacitinib 15 mg QD exposure would still be evaluated against the baseline defined based on the first dose of Upadacitinib 30 mg QD.

In the evaluation of potentially clinically significant laboratory values, the baseline value will be determined by the last non-missing measurement recorded on or before the date of the first dose of study drug in the corresponding treatment group (which may be different than the first dose of study drug in the study). For example, for a subject who started on MTX and switched to upadacitinib 15 mg QD, lab values under upadacitinib 15 mg QD exposure would be evaluated against the baseline value defined as the last non-missing measurement recorded on or before the date of the first dose of upadacitinib 15 mg QD.

A listing of all subjects with any laboratory determination meeting OMERACT criteria of Grade 3 or 4 will be provided by Grade. For creatine phosphokinase and creatinine, NCI CTC criteria will be used. Only subjects with worsening in grade compare to baseline grade will be captured. For each of these subjects, the whole course of the respective parameter will be listed.

#### 9.3.3.3 Assessment of Liver Elevations

The frequencies and percentages of subjects with post baseline liver- specific function test values that meet the criteria of potential clinical interest (as described in Section 9.3.2.4) will be summarized by the actual treatment received at the time of the event occurrence. Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 QD. The treatment exposure groups for



summarizing liver elevations are the same as the ones for long-term AE analysis as described in Section 8.1 and Section 0.

A subject can be counted under different treatment groups if he/she switched treatment and experienced potentially clinical significant laboratory values under different treatment groups.

A listing of potentially clinically significant liver elevations based on criteria specified above will be provided. For each of these subjects, the whole course of the respective parameter will be listed.

### 9.4 Analysis of Vital Signs

### 9.4.1 Variables and Criteria Defining Abnormality

Vital sign variables include sitting systolic blood pressure, sitting diastolic blood pressure, pulse rate, respiratory rate, body temperature, and weight. The criteria for potentially clinically significant vital sign findings are presented in Table 11.

Table 11. Criteria for Potentially Clinically Significant Vital Sign Findings

| Vital Sign | Category | Criteria for Potential Clinically Significant Vital Signs |
|---|---|---|
| Systolic blood pressure | Low | Value $\leq 90$ mmHg and decrease $\geq 20$ mmHg from Baseline |
| | High | Value $\geq$ 160 mmHg and increase $\geq$ 20 mmHg from Baseline |
| Diastolic blood pressure | Low | Value $\leq 50$ mmHg and decrease $\geq 15$ mmHg from Baseline |
| | High | Value $\geq 105$ mmHg and increase $\geq 15$ mmHg from Baseline |
| Weight | High | > 7% increase from baseline |
| | Low | > 7% decrease from baseline |

### 9.4.2 Analysis of Vital Signs for Period 1

Analyses of mean change from baseline in continuous vital sign variables which are measured longitudinally will be performed by visits and by the "as treated" treatment groups of Upadacitinib 15 mg QD, Upadacitinib 30 mg QD, and combined MTX groups. For each change from baseline analysis, the following summary statistics will be



presented for each treatment group: sample size, baseline mean, visit mean, and the mean, standard deviation, and median of the changes from baseline. An ANOVA model with treatment as factor, will be used to test statistical significance for the change from baseline mean among different treatment groups.

The number and percentage of subjects meeting the criteria for potentially clinically significant vital sign values will be summarized by "as treated" treatment group and overall.

# 9.4.3 Analysis of Long-Term Vital Signs

Analyses of mean change from baseline in continuous vital signs variables which are measured longitudinally will be performed by visits and by "as treated" treatment group sequences as described in Section 9.1. For each change from baseline analysis, the following summary statistics will be presented for each treatment group: sample size, baseline mean, visit mean, and the mean, standard deviation, and median of the changes from baseline.

Long-Term Vital Sign will also be summarized based on the number and percentage of subjects meeting the criteria for potentially clinical significant vital sign values and by the actual treatment received at the time of the event occurrence. The treatment groups are the same as the ones for long-term AE analysis as described in Section 8.1 and Section 0. In the evaluation of potentially clinically significant vital sign values, the baseline value will be determined by the last non-missing measurement recorded on or before the date of the first dose of study drug in the corresponding treatment group, similarly as described in Section 9.3.3.2. A subject can be counted under different treatment groups if he/she switched treatment and experienced potentially clinical significant laboratory values under different treatment groups.

In the evaluation of potentially clinically significant vital sign values, the baseline value will be determined by the last non-missing measurement recorded on or before the date of



the first dose of study drug in the corresponding treatment group, similarly as described in Section 9.3.3.2.

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 QD. Mean change from baseline in vital signs for subjects who switched from upadacitinib 30 mg QD to 15 mg QD will be censored at the time of dose switch, and mean change from baseline for values post switch will be summarized separately, similarly as described in Section 9.3.3.1. The treatment groups for summarizing potentially clinical significant vital sign values are the same as the ones for long-term AE analysis as described in Section 8.1 and Section 0. For the purpose of evaluating potentially clinical significant vital sign values, for subjects who switched from upadacitinib 30 mg QD to upadacitinib 15 mg QD, baseline is defined based on the first dose of upadacitinib 30 mg QD, similarly as described in Section 9.3.3.2.

A listing of all subjects with any vital sign values meeting the criteria for potentially clinically significant vital signs will be provided. For each of these subjects, the whole course of the respective parameter will be listed.

# 10.0 Summary of Changes

# 10.1 Summary of Changes between the Previous Version and the Current Version

The primary efficacy analysis and Period 1 reporting have been completed under the SAP version 2.0. The current SAP update applies only to future reporting of long-term analysis.

Updated throughout the SAP to align with Protocol Amendment 5, 6 and 7, including handling of dose switch from upadacitinib 30 mg QD to 15 mg QD (hereafter referred to as "dose switch") and change of study length from 240 to 260 weeks.



- 2. Updated Section 6.0 to clarify analysis details and incorporate additional summary of dose switch.
- 3. Updated Section 7.1 study drug exposure groups to accommodate dose switch.
- 4. Updated Section 8.1.1 and Section 8.1.1 to incorporate handling of dose switch for long-term efficacy analysis.
- 5. Updated Section 8.1.2 to describe the missing data handling approach for the additional sensitivity analysis using longitudinal models for long-term efficacy.
- 6. Updated Section 8.3 to incorporate the additional sensitivity analysis for long-term efficacy.
- 7. Added language to clarify analysis details in Section 9.2.1.1, Section 9.2.1.6, Section 9.2.2.1, Section 9.2.2.3, Section 9.3.3.2, and Section 9.4.3.
- 8. Updated Section 9.2.1.6 and Section 9.4.1 to align with the latest upadacitinib AESI definitions in PSSAP V4.0.
- 9. Updated Section 9.1, Section 0, Section 9.3.3.1, Section 9.3.3.2, Section 9.3.3.3 and Section 9.4.3 to incorporate handling of dose switch for long-term safety analysis.
- Added Appendix C to describe analysis accounting for impact of COVID-19 pandemic.
- 11. Added Section 10.0 for summary of changes and Section 11.0 for SAP version history summary.



# 11.0 Version History

# Table 12. SAP Version History Summary

| Version | Date | Summary |
|---|---|---|
| 1.0 | 27 Dec 2016 | Original version (submitted to FDA to gain feedback). |
| 2.0 | 29 Nov 2017 | Updated to incorporate FDA feedback. Version 2.0 was used for the primary analysis. |
| 3.0 | 17 Dec 2020 | Updated to align with Protocol Amendment 5, 6 and 7, including handling of dose switch from upadacitinib 30 mg QD to 15 mg QD and change of study length from 240 to 260 weeks. Included additional sensitivity analysis for long-term efficacy, and analyses due to COVID-19 impact. |


# 12.0 Appendix

Appendix A OMERACT Criteria
Appendix B NCI CTC Criteria

Appendix C Statistical Analysis to Account for Impact of COVID-19 Pandemic



### Appendix A. OMERACT Criteria

#### Rheumatology Common Toxicity Criteria v.2.0

Based on Woodworth TG, et al. Standardizing assessment of adverse effects in rheumatology clinical trials II. Status of OMERACT Drug Safety Working Group May 2006: OMERACT 8. Standardizing Assessment and Reporting of Adverse Effects in Rheumatology Clinical Trials: Enabling Description of Comparative Safety Profiles for Antirheumatic Therapies

| Safety Profiles for Antirheumati | ic Therapies | | | |
|---|---|---|---|---|
| | 1 – Mild Asymptomatic, or transient Short duration (< 1 week) No change in life style No medication or OTC | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve. (may be prescription), Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation, or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent. Multiple meds Hospitalised > 24 hr Study drug discontinued |
| A. Allergic/Immunologic | | | | |
| A1. Allergic reaction/<br>hypersensitivity (includes drug<br>fever) | Transient rash: drug fever < 38°C: transient, asymptomatic bronchospasm | Generalised urticaria responsive<br>to meds; or drug fever > 38°C,<br>or reversible bronchospasm | Symptomatic bronchospasm requiring meds; symptomatic urticaria persisting with meds, allergy related oedema/angioedema | Anaphylaxis,<br>laryngeal/pharyngeal oedema,<br>requiring resuscitation |
| A2. Autoimmune reaction | Seriologic or other evidence of<br>autoimmune reaction, but<br>patient asymptomatic: all organ<br>function normal and no<br>treatment is required<br>(e.g., vitiligo) | Evidence of autoimmune reaction involving a non-essential organ or functions, requiring treatment other than immunosuppressive drugs (e.g., hypothyroidism) | Reversible autoimmune reaction involving function of a major organ or toxicity requiring short term immunosuppressive treatment (e.g., transient colitis or anaemia) | Causes major organ dysfunction, or progressive, not reversible, or requires long-term administration of high dose immunosuppressive therapy |
| A3. Rhinitis (includes sneezing, nasal stuffiness, post-nasal discharge) | Transient, non-prescription meds relieve | Prescription med. required, slow | Corticosteroids or other<br>prescription med. with persistent<br>disabling symptoms such as<br>impaired exercise tolerance | NA |

| A4. Serum sickness | Transient, non-prescription meds relieve | Symptomatic, slow response to meds (e.g., oral corticosteroids) | Prolonged; symptoms only partially relieved by meds; parenteral corticosteroids required | Major organ dysfunction,<br>requires long-term high-dose<br>immunosuppressive therapy |
|---|---|---|---|---|
| A5. Vasculitis | Localised, not requiring treatment; or rapid response to meds; cutaneous | Symptomatic, slow response to meds (e.g., oral corticosteroids) | Generalised, parenteral corticosteroids required or/and short duration hospitalisation | Prolonged, hospitalisation, ischemic changes, amputation |
| B. Cardiac | 1 | | | |
| B1. Arrhythmia | Transient, asymptomatic | Transient, but symptomatic or recurrent, responds to meds | Recurrent/persistent;<br>maintenance prescription | Unstable, hospitalisation required, parenteral meds |
| B2. Cardiac function decreased | Asymptomatic decline in resting ejection fraction by > 10%, but < 20% of baseline value | Asymptomatic decline of resting ejection fraction ≥ 20% of baseline value | CHF responsive to treatment | Severe or refractory CHF |
| B3. Edema | Asymptomatic (e.g., 1 + feet/calves), self-limited, no therapy required | Symptomatic (e.g., 2 + feet/calves), requires therapy | Symptoms limiting function (e.g., 3 + feet/calves, 2 + thighs), partial relief with treatment prolonged | Anasarca; no response to treatment |
| B4. Hypertension (new onset or worsening) | Asymptomatic, transient increase by > 20 mmHg (diastolic) or to > 150/100 if previously normal, no therapy required | Recurrent or persistent increase > 150/100 or by > 10 mmHg (diastolic), requiring and responding readily to treatment | Symptomatic increase > 150/100, > 20 mmHg, persistent, requiring multi agency therapy, difficult to control | Hypertensive crisis |
| B5. Hypotension (without underlying diagnosis) | Transient, intermittent,<br>asymptomatic, orthostatic<br>decrease in blood pressure<br>> 20 mmHg | Symptomatic, without interference with function, recurrent or persistent > 20 mmHg decrease, responds to treatment | Syncope or symptomatic, interferes with function, requiring therapy and sustained medical attention, dose adjustment or drug discontinuation | Shock |

| B6. Myocardial ischaemia | Transient chest pain/ECG changes; rapid relief with nitro | Recurring chest pain, transient<br>ECG ST-T changes; treatment<br>relieves | Angina with infarction, no or minimal functional compromise, reduce dose or discontinue study drug | Acute myocardial infarction, arrthymia or/and CHF |
|---|---|---|---|---|
| B7. Pericarditis/ pericardial effusion | Rub heard, asymptomatic | Detectable effusion by<br>echocardiogram, symptomatic<br>NSAID required | Detectable on chest x-ray,<br>dyspnoea; or pericardiocentesis;<br>requires corticosteroids | Pulsus alternates with low cardiac output; requires surgery |
| B8. Phlebitis/thrombosis/<br>Embolism (excludes injection<br>sites) | Asymptomatic, superficial, transient, local, or no treatment required | Symptomatic, recurrent, deep vein thrombosis, no anticoagulant therapy required | Deep vein thrombosis requiring anticoagulant therapy | Pulmonary embolism |
| C. General (Constitutional) | | | 1 | |
| C1. Fatigue/malaise (asthenia) | Increase over baseline; most usual daily functions maintained, short term | Limits daily function intermittently over time | Interferes with basic ADL, persistent | Unable to care for self, bed or wheelchair bound > 50% of day debilitating, hospitalisation |
| C2. Fever (pyrexia) (note: fever due to drug allergy should be coded as allergy) | Transient, few symptoms 37.7 – 38.5°C | Symptomatic, recurrent 38.6 – 39.9°C. Relieved by meds | ≥ 40°C; ≤ 24 h, persistent symptoms; partial response to meds | ≥ 40°C, debilitating, > 24 h, hospitalisation; no relief with meds |
| C3. Headache | Transient or intermittent, no meds or relieved with OTC | Persistent, recurring, non-<br>narcotic analgesics relieve | Prolonged with limited response to narcotic medicine | Intractable, debilitating, requires parenteral meds |
| C4. Insomnia | Difficulty sleeping, short term, no interfering with function | Difficulty sleeping interfering with function, use of prescription med | Prolonged symptoms, with limited response to narcotic meds | Debilitating, hospitalisation; no relief with meds |
| C5. Rigors, chills | Asymptomatic, transient, no meds, or non-narcotic meds relieve | Symptomatic, narcotic meds relieve | Prolonged symptoms, with limited response to narcotic meds | Debilitating, hospitalisation; no relief with meds |
| C6. Sweating (diaphoresis) | Episodic, transient | Frequent, short term | Frequent, drenching, disabling | Dehydration, requiring IV fluids/hospitalization > 24 hrs |
| C7. Weight gain | 5% – 9.9% | 10% – 19.9% | 20% – 30% | NA |
| C8. Weight loss | 5% - 9.9% | 10% – 19.9% | 20% – 30% | NA |

| D. Dermatologic | D. Dermatologic | | | |
|---|---|---|---|---|
| D1. Alopecia | Subjective, transient | Objective, fully reversible | Patchy, wig used, partly reversible | Complete, or irreversible even if patchy |
| D2. Bullous eruption | Localised, asymptomatic | Localised, symptomatic, requiring treatment | Generalised, responsive to treatment; reversible | Prolonged, generalised, or requiring hospitalisation for treatment |
| D3. Dry skin | Asymptomatic, controlled with emollients | Symptoms eventually (1 – 2 wks) controlled with emollients | Generalised, interfering with ADL > 2 wks, persistent pruritis, partially responsive to treatment | Disabling for extended period,<br>unresponsive to ancillary<br>therapy and requiring study drug<br>discontinuation for relief |
| D4. Injection site reaction | Local erythema, pain, pruritis, < few days | Erythema, pain, oedema, may include superficial phlebitis, 1 – 2 wks | Prolonged induration, superficial ulceration; includes thrombosis | Major ulceration necrosis requiring surgery |
| D5. Petechiae (without vasculitis) | Few, transient asymptomatic | Dependent areas, persistent up to 2 wks | Generalised, responsive to treatment; reversible | Prolonged, irreversible, disabling |
| D6. Photosensitivity | Transient erythema | Painful erythema and oedema requiring topical treatment | Blistering or desquamation, requires systematic corticosteroids | Generalised exfoliation or hospitalisation |
| D7. Pruritis | Localised, asymptomatic, transient, local treatment | Intense, or generalised, relieved by systematic medication | Intense or generalised; poorly controlled despite treatment | Disabling, irreversible |
| D8. Rash (not bullous) | Erythema, scattered<br>macular/popular eruption;<br>pruritis transient; TOC or no<br>meds | Diffuse macular/popular<br>eruption or erythema with<br>pruritus; dry desquamation;<br>treatment required | Generalised, moist<br>desquamation, requires systemic<br>corticosteroids; responsive to<br>treatment; reversible | Exfoliative or ulcerating; or requires hospitalisation; or parenteral corticosteroids |
| D9. Induration/fibrosis/<br>Thickening (not sclerodermal) | Localized, high density on palpation, reversible, no effect on ADL and not disfiguring | Local areas < 50% body surface,<br>not disfiguring, transient<br>interference with ADL,<br>reversible | Generalized, disfiguring, interferes with ADL, reversible | Disabling, irreversible, systemic symptoms |

| E. Ear/Nose/Throat | | | | |
|---|---|---|---|---|
| E1. Hearing loss | Transient, intermittent, no interference with function | Symptomatic, treatment required, reversible | Interferes with function; incomplete response to treatment | Irreversible deafness |
| E2. Sense of smell | Slightly altered | Markedly altered | Complete loss, reversible | Complete loss, without recovery |
| E3. Stomatitis | Asymptomatic | Painful, multiple, can eat | Interferes with nutrition, slowly reversible | Requires enteral support; residual dysfunction |
| E4. Taste disturbance (dysgeusia) | Transiently altered; metallic | Persistently altered; limited effect on eating | Disabling, effect on nutrition | NA |
| E5. Tinnitus | Intermittent, transient, no interference with function | Requires treatment, reversible | Disabling, or associated with hearing loss | Irreversible deafness |
| E6. Voice changes (includes hoarseness, loss of voice, laryngitis) | Intermittent hoarseness, able to vocalise | Persistent hoarseness, able to vocalise | Whispered speech, slow return of ability to vocalise | Unable to vocalize for extended |
| E7. Xerostomia (dry mouth) | Transient dryness | Relief with meds | Interferes with nutrition, slowly reversible | Extended duration interference with nutrition, requires parenteral nutrition |
| F. Eye/Ophthalmologic | | | | |
| F1. Cataract | Asymptomatic, no change in vision, non-progressive | Symptomatic, partial visual loss, progressive | Symptoms impairing function, vision loss requiring treatment, including surgery | NA |
| F2. Conjunctivitis | Asymptomatic, transient, rapid response to treatment | Symptomatic, responds to treatment, changes not interfering with function | Symptoms prolonged, partial response to treatment, interferes with function | NA |
| F3. Lacrimation increased (tearing, watery eyes) | Symptoms not requiring treatment, transient | Symptomatic, treatment required, reversible | Unresponsive to treatment with major effect on function | NA |
| F4. Retinopathy | Asymptomatic, non-progressive, no treatment | Reversible change in vision; readily responsive to treatment | Disabling change in vision ophthalmological findings reversible, sight improves over time | Loss of sight |

| F5. Vision changes (e.g., blurred, photophobia, night blindness, vitreous floaters) | Asymptomatic, transient, no treatment required | Symptomatic, vision changes not interfering with function, reversible | Symptomatic, vision changes interfering with function | Loss of sight |
|---|---|---|---|---|
| F6. Xerophtalmia (dry eyes) | Mild scratchiness | Symptomatic without interfering with function, requires artificial tears | Interferes with vision/function, corneal ulceration | Loss of sight |
| G. Gastrointestinal | | | | |
| G1. Anorexia | Adequate food intake, minimal weight loss | Symptoms requiring oral nutritional supplementation | Prolonged, requiring iv support | Requires hospitalization for nutritional support |
| G2. Constipation | Asymptomatic, transient, responds to stool softener, OTC laxatives | Symptomatic, requiring prescription laxatives, reversible | Obstipation requiring medical intervention | Bowel obstruction. Surgery required |
| G3. Diarrhea | Transient, increase of 2 – 3 stools/day over pre-treatment (no blood or mucus), OTC agents relieve | Symptomatic, increase 4 – 6 stools/day, nocturnal stools, cramping, requires treatment with prescription meds | Increase > 6 stools/day,<br>associated with disabling<br>symptoms, e.g., incontinence,<br>severe cramping, partial<br>response to treatment | Prolonged, dehydration,<br>unresponsive to treatment,<br>requires hospitalization |
| G4. Dyspepsia (heartburn) | Transient, intermittent, responds to OTC antacids, H-2 blockers | Prolonged, recurrent, requires prescription meds, relieved by meds | Persistent despite treatment,<br>interferes with function,<br>associated with GI bleeding | NA |
| G5. GI bleed (gastritis, gastric or duodenal ulcer diagnosed-define aetiology) | Asymptomatic, endoscopic finding, haemocult + stools, no transfusion, responds rapidly to treatment | Symptomatic, transfusion ≤ 2 units needed; responds to treatment | Haematemesis, transfusion 3 – 4 units, prolonged interference with function | Recurrent, transfusion > 4 units, perforation, requiring surgery, hospitalisation |
| G6. Haematochezia (rectal bleeding) | Haemorrhodial, asymptomatic, no transfusion | Symptomatic, transfusion ≤ 2 units, reversible | Recurrent, transfusion > 3 – 4 units | > 4 units, hypotension, requiring hospitalization |
| G7. Hepatitis | Laboratory abnormalities, asymptomatic, reversible | Symptomatic laboratory<br>abnormalities, not interfering<br>with function, slowly reversible | Laboratory abnormalities persistent > 2 wks, symptoms interfere with function | Progressive, hepato-renal, anasarca, pre-coma or coma |

| G8. Nausea, or nausea/vomiting (use diagnostic term) | Transient, intermittent, minimal interference with intake, rapid response to meds | Persistent, recurrent, requires prescription meds, intake maintained | Prolonged, interferes with daily function and nutritional intake, periodic iv fluids | Hypotensive, hospitalization, parenteral nutrition, unresponsive to out-patient management |
|---|---|---|---|---|
| G9. Pancreatitis | Anylase elevation, intermittent nausea/vomiting, transient, responds rapidly to treatment | Amylase elevation with abdominal pain, nausea, occasional vomiting, responsive to treatment | Severe, persistent abdominal pain with pancreatitic enzyme elevation, incomplete or slow response to treatment | Complicated by shock,<br>haemorrhage (acute circulatory<br>failure) |
| G10. Proctitis | Perianal pruritus, haemorrhoids<br>(new onset), transient, or<br>intermittent, relieved by OTC<br>meds | Tenesmus or ulcerations, anal fissure, responsive to treatment, minimal interference with function | Unresponsive to treatment,<br>marked interference with<br>function | Mucosal necrosis with<br>haemorrhage, infection, surgery<br>required |
| H. Musculoskeletal | | | | |
| H1. Avascular necrosis | Asymptomatic MRI changes, non-progressive | MRI changes and symptoms responsive to rest and analgesia | MRI changes, symptoms requiring surgical intervention | Wheelchair bound; surgical repair not possible |
| H2. Arthralgia | Intermittent transient symptoms, no meds or relieved by OTC meds | Persistent or recurrent symptoms, resolve with meds, little effect on function | Severe symptoms despite meds impairs function | Debilitating, hospitalisation required for treatment |
| H3. Leg cramps | Transient, intermittent, does not interfere with function | Recurrent symptoms, minimally interferes with function or sleep, responds to meds | Persistent, prolonged<br>interference with function or<br>sleep, partial or no response to<br>meds | NA |
| H4. Myalgia | Occasional; does not interfere with function | Frequent, requires meds (non-<br>narcotic); minor effects on<br>function | Major change in function/lifestyle, narcotic pain meds | Debilitating, profound<br>weakness, requires wheelchair,<br>unresponsive to meds |
| I. Neuropsychiatric | | | | |
| I1. Anxiety or Depression (mood alteration) | Symptomatic, does not interfere with function; no meds | Frequent symptoms, responds to meds; interferes with ADL at times | Persistent, prolonged symptoms, partial or no response to meds, limits daily function | Suicidal ideation or danger to self |

| I2. Cerebrovascular ischaemia | NA | Single transient ischaemic event, responsive to treatment | Recurrent transient ischaemic events | Cerebrovascular vascular accident with permanent disability |
|---|---|---|---|---|
| I3. Cognitive disturbance | Subjective symptoms, transient, intermittent, not interfering with function | Objective symptoms, persisting, interferes with daily function occasionally | Persistent, or worsening objective symptoms; interferes with routine daily routine | Debilitating/disabling and permanent; toxic psychosis |
| I4. Depressed consciousness (somnolence) | Observed, transient, intermittent, not interfering with function | Somnolence or sedation, interfering with function | Persistent, progressive, obundation, stupor | Coma |
| I5. Inability to concentrate | Subjective symptoms, does not interfere with function | Objective findings, interferes with function | Persistent, prolonged objective findings or organic cause | NA |
| I6. Insomnia (in absence of pain) | Occasional difficulty sleeping, transient intermittent, not interfering with function | Recurrent difficulty sleeping;<br>requires meds for relief;<br>occasional interference with<br>function | Persistent or worsening difficulty sleeping; severely interferes with routine daily function | NA |
| I7. Libido decreased | Decrease in interest | Loss of interest; influences relationship | Persistent, prolonged interfering with relationship | NA |
| I8. Peripheral motor neuropathy | Subjective or transient loss of deep tendon reflexes; function maintained | Objective weakness, persistent, no significant impairment of daily function | Objective weakness with substantial impairment of function | Paralysis |
| I9. Peripheral sensory<br>neuropathy (sensory<br>disturbance) | Subjective symptoms without objective findings, transient, not interfering with function | Objective sensory loss,<br>persistent, not interfering with<br>function | Prolonged sensory loss or paraethesias interfering with function | NA |
| I10. Seizure | NA | Recurrence of old seizures, controlled with adjustment of medication | Recurrence/exacerbation with partial response to medication | Recurrence not controlled, requiring hospitalization; new seizures |
| I11. Vertigo (dizziness) | Subjective symptoms, transient, intermittent, no treatment | Objective findings, recurrent,<br>meds relieve, occasionally<br>interfering with function | Persistent, prolonged, interfering with daily function; partial response to medication | Debilitating without response to medication, hospitalization |

| J. Pulmonary | | | | |
|---|---|---|---|---|
| J1. Asthma | Occasional wheeze, no interference with activities | Wheezing, requires oral meds, occasional interference with function | Debilitating, requires nasal O <sub>2</sub> | Requires ventilator assistance |
| J2. Cough | Transient, intermittent, occasional OTC meds relieve | Persistent, requires narcotic or other prescription meds for relief | Recurrent, persistent coughing spasms without consistent relief by meds, interferes with function | Interferes with oxygenation; debilitating |
| J3. Dyspnea | Subjective, transient, no interference with function | Symptomatic, intermittent or recurring, interferes with exertional activities | Symptomatic during daily routine activities, interferes with function, treatment with intermittent nasal O <sub>2</sub> relieves | Symptomatic at rest,<br>debilitating, requires constant<br>nasal O <sub>2</sub> |
| J4. Pleuritic pain (pleurisy) | Transient, intermittent symptoms, no treatment or OTC meds relieve | Persistent symptoms, requires prescription meds for relief | Prolonged symptoms, interferes with function, requires frequent narcotic pain relief | Debilitation, requiring hospitalisation |
| J5. Pneumonitis (pulmonary infiltrates) | Asymptomatic radiographic changes, transient, no treatment required | Symptomatic, persistent, requiring corticosteroids | Symptomatic, requiring treatment including O <sub>2</sub> | Debilitating, not reversible; or requiring assisted ventilation |
| J6. Pulmonary function<br>decreased (FVC or carbon<br>monoxide diffusion capacity –<br>DLCO) | 76% – 90% of pre-treatment value | 51% – 75% of pre-treatment value | 26% – 50% of pre-treatment value | ≤ 25% of pre-treatment value |
| Laboratory Data | | | | |
| K. Haematology | | | | |
| K1. Hgb (g/dl) decrease from pre-treatment | 1.0 – 1.4 | 1.5 – 2.0 | 2.1 - 2.9, or Hgb $< 8.0$ , $> 7.0$ | $\geq$ 3.0; or Hgb < 7.0 |
| K2. Leukopenia (total WBC) × 1000 | 3.0 – 3.9 | 2.0 – 2.9 | 1.0 – 1.9 | < 1.0 |
| K3. Neutropenia (× 1000) | 1.5 – 1.9 | 1.0 – 1.4 | 0.5 – 0.9 | < 0.5 |
| K4. Lymphopenia (× 1000) | 1.5 – 1.9 | 1.0 – 1.4 | 0.5 – 0.9 | < 0.5 |



| K5. Platelets (× 1000) | 75 – LLN | 50 – 74.9 | 20 – 49.9; platelet transfusion required | < 20; recurrent platelet transfusions |
|---|---|---|---|---|
| L. Chemistry | | | | |
| L1. Hypercalcaemia (mg/dl) | 1.1 × ULN – 11.5 | 11.6 – 12.5 | 12.6 – 13.5; or symptoms present | > 13.5; or associated coma |
| L2. Hyperglycemia (mg/dl)<br>Fasting | 140 – 160 | 161 – 250 | 251 – 500 | > 500, or associated with ketoacidosis |
| L3. Hyperkalaemia (mmol/l)*** | 5.5 – 5.9 | 6.0 – 6.4 | 6.5 – 7.0 or any ECG change | > 7.0 or any arrhythmia |
| L5. Hypocalcaemia (mg/dl) | 0.9 × LLN – 7.8 | 7.7 – 7.0 | 6.9 – 6.5; or associated with symptoms | < 6.5 or occurrence of tetany |
| L6. Hypoglycemia (mg/dl) | 55 – 64 (no symptoms) | 40 – 54 (or symptoms present) | 30 – 39 (symptoms impair function) | < 30 or coma |
| L7. Hyponatraemia (mmol/l)*** | - | 125 – 129 | 120 – 124 | < 120 |
| L8. Hypokalaemia (mg/dl)*** | - | 3.0 – 3.4 | 2.5 – 2.9 | < 2.5 |
| L9. CPK (also if polymyositis-disease | 1.2 – 1.9 × ULN | 2.0 – 4.0 × ULN | 4.0 × ULN with weakness but<br>without life-threatening signs or<br>symptoms | > 4.0 × ULN with signs or<br>symptoms of rhabdomyolysis or<br>life-threatening |
| L10. Serum uric acid | 1.2 – 1.6 × ULN | $1.7 - 2.9 \times ULN$ | $3.0 - 5.0 \times \text{ULN or gout}$ | NA |
| L11. Creatinine (mg/dl) | 1.1 – 1.3 × ULN | 1.4* – 1.8 × ULN | 1.9 – 3.0 × ULN | > 3.0 × ULN |
| L12. SGOT (AST) | 1.2 – 1.5 × ULN | $1.6 - 3.0 \times ULN$ | 3.1 – 8.0 × ULN | > 8.0 × ULN |
| L13. SGPT (ALT) | 1.2 – 1.5 × ULN | 1.6 – 3.0 × ULN | 3.0 – 8.0 × ULN | > 8.0 × ULN |
| L14. Alkaline phosphatase | 1.1 – 1.5** × ULN | $1.6 - 3.0 \times ULN$ | $3.0-5.0 \times ULN$ | > 5.0 × ULN |
| L15. T. bilirubin | 1.1 – 1.4 × ULN | 1.5 – 1.9 × ULN | 2.0 – 3.0 × ULN | > 3.0 × ULN |
| L16. LDH | 1.3 – 2.4 × ULN | 2.5 – 5.0 × ULN | 5.1 – 10 × ULN | > 10 × ULN |



| M. Urinalysis | M. Urinalysis | | | |
|---|---|---|---|---|
| M1. Haematuria | Micro only | Gross, no clots | Clots, transfusion < 2 units | Transfusion required |
| M2. Proteinuria (per 24 h) | 300 – 500 mg (tr/1+) | 501 – 1999 mg (2+) | 2 – 5.0 g (3+) nephrotic syndrome | 5.0 g (4+) anasarca |
| M3. WBC in urine | NA | NA | Indicating acute interstitial nephritis | Associated with acute renal failure |
| M4. Uric acid crystals | Present without symptoms | NA | With stones or symptoms of stones (e.g., renal colic) | Causing renal outflow obstruction and hospitalization |

<sup>\*</sup> in L11,  $1.5 - 1.8 \times ULN$  is changed to  $1.4 - 1.8 \times ULN$ .

<sup>\*\*</sup> in L14,  $1.1 - 2.0 \times ULN$  is changed to  $1.1 - 1.5 \times ULN$ .

<sup>\*\*\*</sup> in L3, L7 and L8, mg/dl is changed to mmol/l.



## Appendix B. NCI CTC Criteria

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| CPK | $> 1.0 - 2.5 \times ULN$ | $> 2.5 - 5.0 \times ULN$ | > 5.0 – 10.0 × ULN | > 10.0 × ULN |
| Creatinine | > 1.0 – 1.5 × baseline;<br>> 1.0 – 1.5 × ULN | > 1.5 – 3.0 × baseline;<br>> 1.5 – 3.0 × ULN | > 3.0 × baseline;<br>> 3.0 – 6.0 × ULN | > 6.0 × ULN |



#### **Appendix C.** Statistical Analysis to Account for Impact of COVID-19 Pandemic

#### Overview

The COVID-19 pandemic is interfering with the conduct of many ongoing trials, with potential impacts on treatment duration and collection, analysis and the interpretation of clinical trial data. Some protocol-specified visits in the clinical trials may be impacted due to COVID-19 infection or logistical restrictions during the pandemic. For example, some scheduled visits may be missed due to self-quarantine or local government restrictions on travel; some visits may also be delayed or canceled due to healthcare resource constraints during the pandemic. Impacted visits due to COVID-19 will be recorded in the database.

This appendix describes the additional analyses and updates to existing analyses due to COVID-19 impact. At the time of COVID-19 pandemic, all study subjects are in Period 2 of the study. The primary efficacy analysis and Period 1 reporting have been completed in 2017 and are not affected by the COVID-19 pandemic. The analyses described in this appendix are only applicable to Period 2 and future reporting of the long-term analyses.

## **Patient Disposition**

Period 2 patient disposition and reason for discontinuation will be summarized as described in Section 7.0. For subjects who prematurely discontinued study drug or study participation, the reasons for discontinuation will be summarized with two additional categories capturing discontinuation due to COVID-19 infection or logistical restrictions related to the COVID-19 pandemic (as collected in CRF):

- Adverse event (AE)
- Withdrew consent
- Lost to follow-up
- Lack of efficacy
- COVID-19 infection
- COVID-19 logistical restrictions



#### Other

In addition, the number and percentage of subjects with scheduled study visits affected by COVID-19 pandemic will be summarized by treatment group sequences. The impact on study visits will be summarized by the following categories (as collected in CRF) by visit:

- Missed visit
- Virtual visit
- In person, partial assessments done

### **Long Term Efficacy Analysis**

Missing data could occur due to various reasons, including missing visits/assessments, early withdrawal from the study, or missing due to COVID-19 infection or logistic restriction. The probability of having missed visits and missing data due to COVID-19 infection or logistical restrictions related to the COVID-19 pandemic can be reasonably assumed to be unrelated to the unobserved values. Therefore, for the purpose of statistical analysis, it is reasonable to assume that these missing data are missing at random (MAR) and the statistical models that require MAR assumption are appropriate.

As described in Section 9.2.1, longitudinal analysis models MMRM and GLMM will be used for long term efficacy analysis and will be maintained for long term efficacy analysis in the presence of missing data due to COVID-19.

### **Safety Analysis**

In listings of adverse events and deaths, a flag indicating whether the event or death was related to COVID-19 infection will be presented. A listing of COVID-19 related adverse events may be provided.



## 13.0 References

1. Bretz F, Maurer W, Brannath W, et al. A graphical approach to sequentially rejective multiple test procedures. Stats Med. 2009;28(4):586-604.